## FRESENIUS KABI USA, LLC

## STATISTICAL ANALYSIS PLAN

Device:

**AMICUS Separator** 

Clinical Study Protocol:

AMIC-003-CMD

Study Title:

Evaluation of the AMICUS Red Blood Cell Exchange (RBCx)

System in Sickle Cell Patients

Version Date:

21 Feb 2018

| TABLE O | F CONTENTS | PAGE |
|----------|---------------------------------------------------------|------|
| 1 Study | Design | 6 |
| 1.1 S | tudy Objectives | 6 |
| 1.2 S | tatistical Hypothesis | 7 |
| 2 Statis | tical Methodology | 7 |
| 2.1 S | ample Size Calculation | 7 |
| 2.2 A | analysis Population | 8 |
| 2.2.1 | All Subjects Enrolled Population | 8 |
| 2.2.2 | Intent-to-Treat Subjects Population | 8 |
| 2.2.3 | Evaluable Population | 8 |
| 2.3 N | Methods of Statistical Analysis | 10 |
| 3 Analy | ysis Parameters | 10 |
| 3.1 F | rimary Efficacy Parameters | 11 |
| 3.2 S | Secondary Outcome Parameters | 11 |
| 3.3 S | Subject and Procedure Parameters | 12 |
| 3.3.1 | Procedure Selection (CRF 1) | 12 |
| 3.3.2 | Inclusion/Exclusion Criteria and Eligibility (CRF 2, 3) | 13 |
| 3.3.3 | Demographics (CRF 4) | 13 |
| 3.3.4 | Routine Pre-procedure Testing Data (CRF 5) | 13 |
| 3.3.5 | Subject Evaluations Parameters (CRF 5) | 13 |
| 3.3.6 | Subject Laboratory Analysis Parameters (CRF 6) | 14 |
| 3.4 | Concomitant Medications (CRF 7) | 14 |
| 3.5 | Procedure Parameters | 14 |
| 3.5.1 | Procedure Evaluations (CRF 8 & 9) | 14 |

| | 3.5. | .2 Adverse Events (CRF 10 and 21) | 15 |
|---|---|---|---|
| | 3.5. | .3 Adverse Events Post-procedure Assessment (CRF 20) | 15 |
| | 3.5. | .4 Procedure Parameters –Pre-procedure (CRF 11) | 16 |
| | 3.5. | .5 Procedure Parameters –End of Depletion Phase (CRF 12) | 17 |
| | 3.5. | 6.6 Procedure Results (CRF 13) | 17 |
| | 3.5. | 7.7 Replacement RBC Unit Parameters (CRF 14) | 18 |
| | 3.5. | 5.8 Device Alarms (CRF 15) | 18 |
| | 3.5. | Waste Material – RBC Depletion/Exchange (CRF 16) | 18 |
| | 3.5. | 5.10 Waste Material – RBC Exchange (CRF 16) | 19 |
| 2 | 3.6 | Procedure Evaluation and End of Study Parameters (CRF 8, 9 and 17) | 19 |
| 2 | 3.7 | Protocol Deviation (CRF 18) | 20 |
| 4 | Dat | ta Conventions | 20 |
| 4 | 4.1 | Data Collection, Verification, and Monitoring | 20 |
| 4 | 4.2 | Data Handling | 21 |
| | 4.2 | 2.1 Handling of Missing Values | 21 |
| | 4.2 | 2.2 Relative Day Ranges | 21 |
| • | 4.3 | Time and Events Schedule for Study Evaluation Testing Parameters | 21 |
| 5 | Tri | ial Termination Procedures | 21 |
| 6 | Raı | ındomization Schedule | 21 |
| 7 | Sta | atistical References | 21 |
| 8 | Sta | atistical Code for Hypothesis Testing | 21 |
| 9 | Tal | able of Contents for Statistical Output | 22 |
| | 9.1 | Planned Tables <sup>1</sup> | 22 |
| | 9.2 | Planned Listings | 23 |

| Version: | $^{\circ}$ | D-1- | 201 | O |
|----------|------------|------|------|---|
| Wergion: | / 1 | Hen | /111 | 7 |

| STA | TISIT | TCAL | ANAI | VSIS | <b>PLAN</b> |
|-----|-------|------|-------|-----------|-------------|
| OIA | | | AINAI | 7 1 10110 | LLAIN |

# **Evaluation of the AMICUS Red Blood Cell Exchange (RBCx) System in Sickle Cell Patients**

# Signature Page

This Statistical Analysis Plan has been reviewed and approved by the following Fresenius Kabi personnel:

| Hora Ayeni | 02/21/2018 |
|---|---|
| Flora Ayeni, PhD | Date |
| Senior Biostatistician | |
| Clinical Affairs | |
| Jason Friedmann Lead Clinical Research Specialist Clinical Affairs | <u>02 21 2018</u><br>Date |
| Carrie Pineda, MS/MBA Senior Director Clinical Affairs | 02/21/2018<br>Date |

#### 1 STUDY DESIGN

The AMICUS Red Blood Cell Exchange (RBCx) procedure will be evaluated using a multi-center, single-arm, open label study design. Up to a total of 100 subjects meeting all eligibility criteria will be enrolled to complete a minimum of 62 evaluable RBCx procedures.

The RBCx is a type of therapeutic procedure used to remove red blood cells (RBCs) from sickle cell disease (SCD) subjects, exchanging them for healthy donor RBCs and/or crystalloid or colloid solutions to maintain fluid balance. Depending upon the replacement fluid(s) (RF) used, the procedure can be considered an RBC Exchange or an RBC Depletion/Exchange procedure. The RBC Depletion/Exchange procedure is a modification of the RBC Exchange procedure. Removal of RBCs may be performed manually or using an apheresis device. The removal of RBCs and replacement with healthy donor RBCs is most frequently used in the treatment of patients with complications of sickle cell disease. The type of procedure performed (RBC Exchange or RBC Depletion/Exchange) will be prescribed by the physician.

The study will have a lead-in phase for training purposes and the lead-in subjects will not be included in the evaluable population. Evaluable subjects will be obtained in two stages. In the first stage up to 40 subjects 18 years old or older will be enrolled to complete 31 evaluable procedures. An interim report including summary statistics and safety-related data will be reviewed by a Data Safety Monitoring Board (DSMB). The DSMB primary responsibilities are to monitor the safety of the trial participants, to review safety-related data, to evaluate the frequency and severity of adverse events, and to judge the quality and integrity of study data. A separate analysis plan is written for the interim report.

Following the DSMB review the report will be submitted to the FDA for review as an IDE supplement. This supplement must be approved before the start of the second stage of the study. This stage will enroll pediatric subjects 6 to 17 years old.

## 1.1 Study Objectives

The primary objective of the study is to evaluate the accuracy of the subject's original RBCs remaining (Actual FCR) as measured by subject's post-procedure Hb S at the end of the procedure to the Target FCR.

The secondary objectives are:

- To evaluate the accuracy of subject hematocrit (Hct) post-procedure (End Hct)
- To evaluate subject cellular loss (white blood cells, platelets) post-procedure
- To evaluate the cellular content of the waste material

 To evaluate device related serious adverse events during the procedure and approximately 18 to 24 hours post-procedure

#### 1.2 Statistical Hypothesis

Hypothesis testing will be performed to evaluate the primary objective of the 95% confidence interval around the mean ratio of actual to target FCR as measured by Hb S in the subjects pre- and post-procedure to a pre-defined FCR range of 0.75 to 1.25.

The primary hypothesis set for the 2-sided test is given as:

H<sub>0</sub>: P<sub>T</sub> LL<0.75 and/or P<sub>T</sub> UL>1.25

Versus

 $H_1: 0.75 \le LL P_T UL \le 1.25$ 

Where  $P_T$  = the 95% CI for AMICUS mean ratio; LL = Lower limit; and UL = Upper limit.

We will reject  $H_0$  at the alpha level of significance if the entire 95% confidence interval around the mean ratio is within the predefined range. Stated explicitly, if the lower limit of the 95% confidence interval around the mean ratio is greater than or equal to the lower predefined range boundary (0.75) and simultaneously the upper limit of the 95% confidence interval around the mean ratio is less than or equal to the upper predefined range boundary (1.25).

Hypothesis testing is not planned for secondary objectives. Summary statistics (mean, standard deviation, minimum, median, maximum, and count) of the RBC Exchange and RBC Depletion/Exchange procedure data will be used to evaluate the secondary objectives: evaluation of the accuracy of subject End Hct, accuracy of Fluid Balance, subject cellular loss post-procedure, and serious device related adverse events.

Hypothesis testing is not planned for the interim report. Summary statistics (mean, standard deviation, minimum, median, maximum, and count) of the RBC Exchange and RBC Depletion/Exchange procedure data will be used to evaluate the primary and secondary objectives.

## 2 STATISTICAL METHODOLOGY

#### 2.1 Sample Size Calculation

The sample size needed for the study design is given as:

$$N=2(Z_1-\alpha+Z_1-\beta)^2 \sigma^2 \div \delta^2$$

Where  $Z_1$ - $\alpha$  and  $Z_1$ - $\beta$  are the standard normal deviates corresponding to 1 minus significance level ( $\alpha$ ) and 1 minus the type II error ( $\beta$ ) respectively,  $\sigma^2$  is the variance or squared standard deviation of the outcome and  $\delta$  is the margin.

Since we planned to have a 90% power at the 0.025 significance level to detect equivalence to a ratio of 1, then the sample size with the margin of 0.25 and observed standard deviation of the difference of 0.43 with  $\beta$  =0.10 will yield:

$$N = 2(1.96 + 1.28)^2 \cdot 0.43^2 \div .25^2 = 2(10.4976) \cdot 0.185 \div 0.0625 = 62.$$

Therefore, a sample size of 62 evaluable procedures will be used to demonstrate that AMICUS is within a margin of 25% with at least 95% (2-sided) confidence and at least 90% power.

## 2.2 Analysis Population

## 2.2.1 All Subjects Enrolled Population

The All Subjects Enrolled population will consist of those subjects who signed an informed consent. The safety population will consist of all enrolled subjects.

## 2.2.2 Intent-to-Treat Subjects Population

The Intent-to-Treat population will consist of those enrolled subjects who successfully complete the AMICUS Separator procedures, and exclude subjects who participated in a Lead-in procedure.

#### 2.2.3 Evaluable Population

The Evaluable population will consist of those enrolled subjects who successfully complete the AMICUS Separator procedures, have values reported for parameters required to calculate the primary endpoint (e.g., day of procedure pre- and post-procedure Hb S results are obtained) and the evaluability criteria are met. These are circumstances during or associated with a RBCx procedure that may cause the primary or secondary endpoint to be non-evaluable. These are stated in Section 13.6 of the protocol. Primary and secondary objectives will be evaluated using the Evaluable population.

If the data required for determining the evaluability of this population is missing, the subject will be non-evaluable. Reasons for non-evaluability of this population will be revisited by the Sponsor prior to database lock. If additional reasons for non-evaluability are identified at this time, all affected statistical documents and SAS programs will be updated accordingly.

# **Evaluability Criterion 1: Procedure Completion**

This Criterion indicates whether or not subjects have a completed collection procedure.

**Evaluability Criterion 2:** If reinfusion was performed, post-procedure blood sample must be taken prior to reinfusion.

Evaluability Criterion 3: Did operator change subject HCT, Avg RF Hct or Total Blood Volume after procedure start

## **Evaluability Criterion 4: Average RF Hct Accuracy**

This Criterion indicates If the absolute difference of the Average Replacement Fluid Hematocrit (%) and Calculated Average Replacement Fluid Hematocrit (%) values is less than or equal to 5 Hematocrit points the calculated A:T FCR Ratio and Calculated End Hct Accuracy are evaluable. If the absolute difference of the Average Replacement Fluid Hematocrit (%) and Calculated Average Replacement Fluid Hematocrit (%) values is less than or equal to 5 Hematocrit points the Calculated A: T FCR Ratio, Calculated Depletion Hct Accuracy and Calculated End Hct Accuracy are evaluable, where Calculated Average Replacement Fluid Hematocrit (%) is equal to the sum of the red cell volume in the RBC units divided by the sum of the total volume in the RBC units. The red cell volume of each unit is defined as the product of the hematocrit and the volume of each individual unit. N is equal to the number RBC units transfused. If the absolute difference of the Average Replacement Fluid Hematocrit (%) and Calculated Average Replacement Fluid Hematocrit (%) values is greater than 5 Hematocrit points then calculated A:T FCR Ratio and Calculated End Hct Accuracy are non-evaluable.

## **Evaluability Criterion 5: Input Hematocrit Difference**

If absolute difference of Subject Hematocrit (%) and Pre-procedure Hematocrit (%) value is less than or equal to 5 Hematocrit points then Calculated A:T FCR Ratio, Calculated Depletion Hct Accuracy and Calculated End Hct Accuracy are evaluable. If absolute difference of Subject Hematocrit (%) and Pre-procedure Hematocrit (%) value is greater than 5 Hematocrit points then Calculated A:T FCR Ratio, Calculated Depletion Hct Accuracy and Calculated End Hct Accuracy are non-evaluable.

#### **Evaluability Criterion 6: Input FCR Difference**

For procedure in which the Fraction of Cells Remaining (%) instead of Replacement Volume (mL) is used to program the inputs, apply the following Evaluability criteria. If the absolute difference of the Fraction of Cells Remaining (%) and Calculated Fraction of Cells Remaining (%) value is less than or equal to 6 percent points then the Calculated A:T FCR Ratio, Calculated Depletion Hct Accuracy and Calculated End Hct are evaluable. If the absolute difference of the Fraction of Cells Remaining (%) and Calculated Fraction of Cells Remaining (%) value is greater than 6 percent points then the Calculated A:T FCR Ratio is not evaluable.

Check if Fraction of Cells Remaining was used as an input. If the following is true then continue on to the evaluability criteria. If the following is not true Fraction of Cells Remaining was not used as an input and the evaluability criterion is not applicable. Note that the evaluability criterion also does not apply if NA is entered for Target Hemoglobin S (%) and/or Actual Hemoglobin S (%).

#### 2.3 Methods of Statistical Analysis

Summary statistics (N, mean, standard deviation, median, minimum, and maximum) will be reported on all continuous (numeric) parameters. Descriptive statistics (e.g., counts and percentages) will be reported on categorical (non-numeric) parameters. All summary statistics will be presented at rounded precision. No estimates will be truncated.

Hypothesis testing will be performed at the conclusion of the study to evaluate the primary objective of 95% confidence interval around the mean ratio of actual to target FCR as measured by Hb S in the subjects' pre- and post-procedure to a pre-defined FCR range of 0.75 to 1.25.

Hypothesis testing will not be performed for the interim analyses and summary statistics will be performed for the Interim report.

All calculations will be performed using SAS 9.4 (Windows platform).

#### 3 ANALYSIS PARAMETERS

All parameters are reported as "[measured]" or "[calculated]". The former indicates that the parameter was collected on a CRF. The latter indicates that the parameter was calculated based on CRF data. The details of all parameter calculations will be provided in the study Algorithms Document.

As a general rule, any parameter values that are censored (left or right) will be analyzed as the numeric version of the observed detection limit (e g, <1.0 will be analyzed as 1.0). The parameters associated with the depletion phase data are only applicable for RBC Depletion/Exchange procedures.

All parameters will be listed for all enrolled subjects. All procedures results summarized will be presented for the evaluable subjects. Summary statistics (mean, standard deviation, minimum, median, maximum, and count) will be presented.

All parameters documented will be available in SAS analysis datasets.

#### 3.1 Primary Efficacy Parameters

The primary efficacy parameter is the subject's original RBCs remaining (Actual FCR) as measured by subject's post-procedure Hb S at the end of the procedure to the target FCR. Hypothesis testing will be performed to evaluate the primary objective of 95% confidence interval around the mean ratio of actual to target FCR as measured by Hb S in the subjects' pre- and post-procedure to a pre-defined FCR 0.75 to 1.25. This parameter will be provided in a listing for the All Enrolled Subjects population.

#### 3.2 Secondary Outcome Parameters

The following secondary objectives will be assessed using the appropriate Evaluable Subject population. The overall procedure subject cellular percent losses, plasma hemoglobin delta, and calculated target End Hct will be calculated. The Exchange procedures and Depletion/Exchange procedures total cell losses, plasma hemoglobin delta, and calculated target End Hct accuracy will be presented.

The waste material for the exchange procedures and Depletion/Exchange procedures will be evaluated for volume, total WBC and platelet counts. For the Depletion/Exchange procedures the depletion phase and exchange phase will be evaluated separately.

#### A. Overall Procedures:

- Subject WBC Percent Loss (%)
- Subject RBC Percent Loss (%)
- Subject Platelet Percent Loss (%)
- Subject Plasma Hemoglobin Delta (mg/dL)
- Calculated Target End Hct Accuracy.

#### B. Exchange Procedures:

- Exchange Procedure Waste Material Volume (mL)
- Exchange Procedure Waste WBC Count (x10<sup>10</sup>)
- Exchange Procedure Waste RBC Count (x10<sup>10</sup>)
- Exchange Procedure Waste Platelet Count (x10<sup>11</sup>)

Calculated Target End Hct Accuracy

Primary and secondary parameters calculations are in the Algorithm Document.

#### C. Depletion/Exchange Procedures:

#### **Depletion Phase**

- Depletion Phase Waste Material Volume (mL)
- Depletion Phase Waste WBC Count (x10<sup>10</sup>)
- Depletion Phase Waste Platelet Count (x10<sup>11</sup>)
- Calculated Depletion Hct Accuracy
- Subject Depletion Phase Plasma Hemoglobin Delta (mg/dL)

## Exchange Phase

- Exchange Phase Waste WBC Count (x10<sup>10</sup>)
- Exchange Phase Waste Platelet Count (x10<sup>11</sup>)
- Calculated Target End Hct Accuracy

## 3.3 Subject and Procedure Parameters

# 3.3.1 Procedure Selection (CRF 1)

The procedure selection parameters to be presented are:

Is this a lead-in procedure? (Yes / No)

- If Yes,
  - Lead-in RBC Exchange
  - Lead-in RBC Depletion Exchange
- If No,
  - RBC Exchange
  - RBC Depletion/Exchange

Listing and summary statistics for all parameters will be reported.

## 3.3.2 Inclusion/Exclusion Criteria and Eligibility (CRF 2, 3)

Listing of all inclusion/exclusion and subject eligibility will be reported.

#### 3.3.3 Demographics (CRF 4)

The demographics parameters to be presented are:

- 1. Date of birth [measured]
- 2. Sex
- 3. Ethnicity
- 4. Race
- 5. Subject age (years) at the time informed consent is obtained.
- 6. Subject age (years) at the time of procedure

Listing and summary statistics for all parameters will be reported.

# 3.3.4 Routine Pre-procedure Testing Data (CRF 5)

The routine pre-procedure testing data to be presented are:

- 1. Sample date (Mmm-dd-yyyy)
- 2. Sample time (hh:mm)
- 3. Actual Hb S (%)
- 4. Target Hb S (%)
- 5. Hct (%)

Listing and summary statistics for all parameters will be reported.

## 3.3.5 Subject Evaluations Parameters (CRF 5)

The subject evaluations parameters to be presented for all procedures are:

- 1. Primary Diagnosis (1=SS, 2=SB-0 thal, 3=SCD, 4=Other (specify))
- 2. Weight (lbs) [measured] [Pre-Procedure]
- 3. Height (in) [measured] [Pre-Procedure]
- 4. Systolic Blood Pressure (mmHg) [measured] [Pre, End of Depletion Phase, and Post-procedure]
- 5. Diastolic Blood Pressure (mmHg) [measured] [Pre, End of Depletion Phase, and Post-procedure]
- 6. Temperature (°F) [measured] [Pre, End of Depletion Phase, and Post-procedure]
- 7. Pulse (bpm) [measured] [Pre, End of Depletion Phase, and Post-procedure]
- 8. Respiration Rate (breaths/min) [measured] [Pre, End of Depletion Phase, and Post-procedure]

Listing and summary statistics for all parameters will be reported.

# 3.3.6 Subject Laboratory Analysis Parameters (CRF 6)

The subject laboratory parameters to be presented are:

- 1. White Blood Cell Count (WBC)  $(x10^3/\mu L)$  [measured] [Pre-procedure, End of Depletion, and Post-procedure]
- 2. Red Blood Cell Count (RBC) ( $x10^6/\mu L$ ) [ measured] ][Pre- procedure, End of Depletion, and Post-procedure]
- 3. Platelet Count  $(x10^3/\mu L)$  [measured] [Pre-procedure, End of Depletion, and Post-procedure]
- 4. Hct (%) [measured] ][Pre- procedure, End of Depletion, and Post-procedure]
- 5. Plasma Hb (mg/dL) [measured] [Pre- procedure, End of Depletion, and Post-procedure
- 6. Hb A (%) [measured] [Pre- and Post-procedure]
- 7. Hb S (%) [measured] [Pre- and Post-procedure]
- 8. Hb C (%) [measured] [Pre- and Post-procedure]
- 9. Hb F (%) [measured] [Pre- and Post-procedure]
- 10. Hb A2 (%) [measured] [Pre- and Post-procedure]
- 11. Pregnancy test [measured] [Pre-procedure]

Listing and summary statistics for all parameters will be reported.

# 3.4 Concomitant Medications (CRF 7)

Concomitant medications used by the subjects for seven days prior to and during the study procedures will be listed in data listings only using the Medical Dictionary for Regulatory Activities (MedDRA) version 18.0 and World Health Organization Drug Dictionary (WHO Drug) version March 2015 dictionaries. No formal summary table will be generated.

#### 3.5 Procedure Parameters

## 3.5.1 Procedure Evaluations (CRF 8 & 9)

The measured procedure evaluation parameters are:

- 1. Procedure Date (Mmm-dd-yyyy)
- 2. End Time (hh:mm)
- 3. Venous Access Used (Peripheral IV, Temporary Catheter, Long Term/Permanent Catheter(Two single lumen ports/One double lumen port)
- 4. Replacement Fluid Used (Saline/Albumin/Custom (specify))
- 5. Anticoagulant Type: (ACD-A/Custom (specify))
- 6. Was reinfusion selected prior to the start of the procedure? (Yes/No)

- 7. Subject Total Sample Volume Removed (mL)
- 8. Custom Prime (Full/Partial/None)
- 9. Was Prime diverted? (Yes/No)
- 10. Was a blood warmer used during the procedure? (Yes/No). If Yes, provide the prime volume (mL)
- 11. Was Saline bolus performed? (Yes/No)
- 12. Was the procedure ended prior to or extended beyond (± 50 mls) of the Target RF Volume? (Yes/No)
- 13. At the end of the procedure, was reinfusion performed? (Yes/No). If Yes, was a sample taken prior to reinfusion? (Yes/No)

Listing and summary statistics for all parameters will be reported.

## 3.5.2 Adverse Events (CRF 10 and 21)

Adverse events (AE) will be recorded through the completion of each Procedure type (during and approximately 18 to 24 hours post procedure). AEs will be presented using MedDRA coding for AEs which requires the site to record the descriptors. Events classified as "Other" will be presented as verbatim terms. An AE type occurring multiple times per subject will be counted once for subject-reported frequencies.

The frequency of subjects who reported AEs and the frequency of AEs reported by and across severity, seriousness, relationship to procedure, and relationship to device will be presented overall, and by site for all subjects enrolled in the study.

Listings and summary tables of AEs/SAEs, and incidence of AEs/SAEs will be reported during the procedure and at post-procedure follow-up of the study.

# 3.5.3 Adverse Events Post-procedure Assessment (CRF 20)

The sites have up to 2 attempts to contact each subject and record the following:

- 1. Was subject contacted on the first attempt? (Yes/No/Not Done).
- 2. Date of first attempt (Mmm-dd-yyyy) / Time of first attempt (hh:mm).
  - a. Was subject contacted on the second attempt? (Yes/No/Not Done).
  - b. Date of second attempt (Mmm-dd-yyyy) / Time of second attempt (hh:mm).
  - c. If No contact by telephone, was a certified letter sent? (Yes/No)
- 3. Was there an AE that occurred during procedure with an outcome of continuing? (Yes/No). If Yes, record all the AE numbers as referenced on the AE page.
- 4. Current outcome of continuing adverse event are:

- a. Recovered (End Date) (Mmm-dd-yyyy)
- b. Recovered with Sequela(e) (End Date) (Mmm-dd-yyyy)
- c. Continuing
- d. Death (Date of Death) (Mmm-dd-yyyy)
- 5. Did the subject experience any AE post-procedure? (Yes/No/Unknown). If Yes, record AE on the AE-post procedure form

Listing of adverse event post-procedure assessment will be reported

## 3.5.4 Procedure Parameters - Pre-procedure (CRF 11)

The procedure parameter results are:

#### Input Parameter

- 1. Fraction Cells Remaining (%)
- 2. End Hct (%)
- 3. Depletion Hct (%)\*
- 4. Replacement Volume (mL)
- 5. Fluid Balance (mL)
- 6. AC Ratio
- 7. Start Prime Hct (%)
- 8. End Prime Hct (%)

#### **Estimator Parameter**

- 1. Whole Blood Flow Rate (mL/min)
- 2. Procedure Time (min)
- 3. Anticoagulant to Subject (mL)
- 4. Anticoagulant Used (mL)
- 5. Other Replacement Fluid (mL)
- 6. Depletion Red Cell Volume (mL)

#### Input Parameter

1. Subject Hct (%)

Was value changed during Procedure? (Yes/No) If Yes Final value-----

2. Average Replacement Fluid Hct (%)

Was value changed during Procedure? (Yes/No) If Yes Final value-----

3. Total Blood Volume (mL)

Was value changed during Procedure? (Yes/No) If Yes Final value-----

- 4. Maximum Whole Blood Flow Rate (mL/min)
  Was value changed during Procedure? (Yes/No) If Yes Final value------
- Citrate Infusion Rate (CIR) (mg/kg/min)
   Was value changed during Procedure? (Yes/No) If Yes Final value------

Listing and summary statistics of all parameters will be reported.

## 3.5.5 Procedure Parameters –End of Depletion Phase (CRF 12)

The end of depletion phase parameter results are:

- 1. Fluid Balance (mL)
- 2. Depletion Hct (%)
- 3. Whole Blood Processed (mL)
- 4. Replacement Fluid Albumin Returned (mL)
- 5. Replacement Fluid Saline Returned (mL)
- 6. Custom Replacement Fluid Returned (mL)
- 7. Plasma Returned (mL)
- 8. Procedure Time (min)
- 9. Anticoagulant Used (mL)
- 10. Anticoagulant to Subject (mL)
- 11. Saline to Subject (mL)

Listing and summary statistics of all parameters will be reported.

## 3.5.6 Procedure Results (CRF 13)

The procedure parameter results are:

- 1. Procedure Time (min)
- 2. Fraction Cells Remaining (%)
- 3. End Hct (%)
- 4. Fluid Balance (mL)
- 5. Red Blood Cell Mass Balance
- 6. Whole Blood Processed (mL)
- 7. Replacement Fluid to Subject (mL)
- 8. Anticoagulant to Subject (mL)
- 9. Anticoagulant Used (mL)
- 10. Saline to Subject (mL)
- 11. Replacement Fluid Albumin Returned (mL)
- 12. Replacement Fluid RBC Returned (mL)

- 13. Replacement Fluid Saline Returned (mL)
- 14. Custom Replacement Fluid Returned (mL)

Listing and summary statistics of all parameters will be reported.

## 3.5.7 Replacement RBC Unit Parameters (CRF 14)

Replacement RBC unit parameters to be presented are:

- 1. Type of RBC Unit
- 2. Unit Identification Number
- 3. Sample Date (Mmm-dd-yyyy)
- 4. Sample Time (hh:mm)
- 5. Hct (%)
- 6. Volume (mL)
- 7. ABO Type/Rh Factor
- 8. Expiration Date
- 9. Plasma Hb (mg/dL)
- 10. Confirmation of Sickle Trait Negative
- 11. Confirmation of Leukoreduction
- 12. Confirmation of Rh(D) compatibility

Listing and summary statistics of all parameters will be reported.

## 3.5.8 Device Alarms (CRF 15)

Device alarms as it occurs during the procedure will be reported with its frequency.

Did alarm(s) occur during the procedure? (Yes/No)

- If yes, record all alarms that occurred and their frequency.

Listings and summary table of all device alarm will be reported by the alarm code, description and frequency.

# 3.5.9 Waste Material – RBC Depletion/Exchange (CRF 16)

The RBC waste material parameters to be presented are:

- 1. Gross Weight (g)
- 2. Tare Weight (g)
- 3. Volume (mL)
- 4. White Blood Cell Count (WBC)  $(x10^3/\mu L)$
- 5. Total WBC Count (x10<sup>9</sup>)

- 6. Platelet Count  $(x10^3/\mu L)$
- 7. Total Platelet Count (x10<sup>11</sup>)
- 8. Hct (%)

Listing and summary statistics of all parameters will be reported.

## 3.5.10 Waste Material – RBC Exchange (CRF 16)

The RBC waste material parameters to be presented are:

- 1. Gross Weight (g)
- 2. Tare Weight (g)
- 3. Volume (mL)
- 4. White Blood Cell Count (WBC)  $(x10^3/\mu L)$
- 5. Total WBC Count (x10<sup>9</sup>)
- 6. Platelet Count  $(x10^3/\mu L)$
- 7. Total Platelet Count (x10<sup>11</sup>)
- 8. Hct (%)

Listing and summary statistics of all parameters will be reported.

# 3.6 Procedure Evaluation and End of Study Parameters (CRF 8, 9 and 17)

The evaluability criteria in section 13.6 of the protocol to be presented are:

- If procedure is terminated prior to completion, the procedure is non-evaluable.
- If reinfusion is performed, the post-procedure blood sample must be drawn prior to reinfusion or it is not evaluable.
- Operator should not change subject Hct, Avg RF Hct, or Total Blood Volume after procedure start or it is not evaluable.
- If a saline bolus is performed, End Hct is not evaluable.

The End of Study parameters to be presented are:

Was the procedure completed? (Yes / No)

- If No, the primary reason will be presented:
  - Adverse Events
  - Venous Access Issue (Non-Adverse Event)
  - Instrument Alarm (specify)
  - Disposable Issue:

- o Leak
- o Kink
- o Misassembly
- o Other
- Hardware Issue
- Investigator Decision
- Subject Decision
- Protocol Deviation/Violation
- Other (please describe)

Listing of all subjects that completed the procedure will be presented and subjects that did not complete the procedure will be reported as per a reason above.

#### 3.7 Protocol Deviation (CRF 18)

Protocol deviations will be presented in data listings only. No formal summary table will be generated.

Listing of protocol deviation will include:

- 1. Was a protocol deviation recorded? (Yes/No)
- 2. Date of the deviation
- 3. Protocol deviation
  - a. Inclusion criteria
  - b. Exclusion criteria
  - c. Sampling /testing issues
  - d. Procedure related issues
  - e. Subject receives wrong treatment or incorrect dose
  - f. Informed consent issues
  - g. Follow-up not performed
  - h. Follow-up outside of window
  - i. Other

#### 4 DATA CONVENTIONS

## 4.1 Data Collection, Verification, and Monitoring

Refer to protocol Section 12, Data Quality Assurance.

#### 4.2 Data Handling

#### 4.2.1 Handling of Missing Values

No missing or incomplete dates will be imputed for this study. No missing or incomplete parameter results will be imputed for this study.

#### 4.2.2 Relative Day Ranges

Not applicable to this study.

# 4.3 Time and Events Schedule for Study Evaluation Testing Parameters

Refer to protocol Section 8.2, Study Procedures/Methodology, Tables 2 to 6.

## 5 TRIAL TERMINATION PROCEDURES

There are no plans for prematurely terminating this study. However, site closure or study termination may be decided at any time by the sponsor or site investigator due to safety concerns, inadequate study subject enrollment, and failure to comply with the study protocol, regulatory requirements, and Good Clinical Practices.

#### 6 RANDOMIZATION SCHEDULE

Not applicable for this study

#### 7 STATISTICAL REFERENCES

Base SAS 9.4 Procedures Guide, Second Edition, Volumes 1-4 (March 2013). SAS Publishing: Cary, NC.

## 8 STATISTICAL CODE FOR HYPOTHESIS TESTING

A SAS macro will be written for generating the applicable output. The macro will be located in the I drive.

# 9 TABLE OF CONTENTS FOR STATISTICAL OUTPUT

# 9.1 Planned Tables<sup>1</sup>

| Table Number | Section | Description of Output |
|---|---|---|
| Table 14.1 | Patients Disposition | Summary of Subjects Disposition (All Subjects Enrolled) |
| Table 14.2.1 | Procedure Evaluability/End of Study | Summary of Procedure Evaluability<br>(Intent-to-Treat Subjects ) |
| Table 14.2.2 | Procedure Selection Parameters<br>Section 3.3.1 | Summary of Procedure Selection Parameters (All Subjects Enrolled) |
| Table 14.3 | Demographic Parameters<br>Section 3.3.3 | Summary of Demographic Parameters (All Subjects Enrolled) |
| Table 14.4 | Routine Pre-procedure Testing Data<br>Section 3.3.4 | Summary of Routine Pre-Procedure Testing Data<br>(Intent-to-Treat Subjects) |
| Table 14.5 | Subject Evaluation Parameters<br>Section 3.3.5 | Summary of Subject Evaluation Parameters (All Subjects Enrolled) |
| Table 14.6 | Subject Laboratory Parameters<br>Section 3.3.6 | Summary of Subject Laboratory Parameters (All Subjects Enrolled) |
| Table 14.7 | Primary Endpoint Parameters<br>Section 3.1 | Analysis of Primary Endpoint Parameters (All Evaluable Subjects) |
| Table 14.8 | Secondary Endpoint Parameters<br>Section 3.2 | Summary of Secondary Endpoint Parameters (All Evaluable Subjects) |
| Table 14.9 | Procedure Evaluation<br>Section 3.5.1 | Summary of Procedure Evaluation Parameters (All Evaluable Subjects) |
| Table 14.10.1 | Adverse Events During the Procedure Section 3.5.2 | Summary of Adverse Events During the Procedure (All Subjects Enrolled) |
| Table 14.10.2 | Adverse Events During the Procedure<br>Section 3.5.2 | Summary of Adverse Events During the Procedure by Site (All Subjects Enrolled) |
| Table 14.10.3 | Incidence of Adverse Events<br>Section 3.5.2 | Incidence of Adverse Events During the Procedure (All Subjects Enrolled) |
| Table 14.10.4 | Incidence of Adverse Events<br>Section 3.5.2 | Incidence of Adverse Events During the Procedure by Site(All Subjects Enrolled) |
| Table 14.11.1 | Adverse Events Post-procedure<br>Section 3.5.2 | Summary of Adverse Events Post-procedure (All Subjects Enrolled) |
| Table 14.11.2 | Adverse Events Post-procedure<br>Section 3.5.2 | Summary of Adverse Events Post-procedure by Site (All Subjects Enrolled) |
| Table 14.11.3 | Incidence of AE Post-procedure<br>Section 3.5.2 | Incidence of Adverse Events Post-procedure (All Subjects Enrolled) |
| Table 14.11.4 | Incidence of AE Post-procedure<br>Section 3.5.2 | Incidence of Adverse Events Post-procedure by Site (All Subjects Enrolled) |
| Table 14.12.1 | Procedure Parameters-Pre-procedure<br>Section 3.5.4 | Summary of Input and Estimator Parameters (All Evaluable Subjects) |
| Table 14.12.2 | Procedure Parameters-End of Depletion Phase<br>Section 3.5.5 | Summary of Procedure Parameters<br>End of Depletion Phase (All Evaluable Subjects) |
| Table 14.13.1 | Procedure Results<br>Section 3.5.6 | Summary of Procedure Results (All Evaluable Subjects) |
| Table 14.13.2 <sup>2</sup> | Procedure Results<br>Section 3.5.6 | Summary of Empirical RBC Mass Balance Excluding Outlier(s) (All Evaluable Subjects) |
| Table 14.14 | Replacement RBC Unit Parameters<br>Section 3.5.7 | Summary of Replacement RBC Unit Parameters (All Evaluable Subjects) |
| Table 14.15 | Device Alarms Section 3.5.8 | Summary of Device Alarms (All Subjects Enrolled) |
| Table 14.16.1 | Waste Material-RBC Depletion/Exchange<br>Section 3.5.9 | Summary of Waste Material-RBC Depletion/Exchange Procedure (All Evaluable Subjects) |
| Table 14.16.2 | Waste Material-RBC Exchange<br>Section 3.5.10 | Summary of Waste Material-RBC Exchange Procedure (All Evaluable Subjects) |
| Table 14.17 | End Hematocrit Section 3.5.4 | Summary of End Hematocrit (All Evaluable Subjects) |

## 9.2 Planned Listings

| Listing Number | Section | Description of Output |
|---|---|---|
| Listing 16.1 | Patients Disposition | Listing of Subjects Disposition (All Subjects Enrolled) |
| Listing 16.2 | Procedure Evaluability/End of Study | Listing of Procedure Evaluability/End of Study (All Subjects Enrolled) |
| Li sting 16.3.1 | Inclusion/Exclusion and Eligibility | Listing of Inclusion Criteria (All Subjects Enrolled) |
| Listing 16.3.2 | Inclusion/Exclusion and Eligibility | Listing of Exclusion Criteria (All Subjects Enrolled) |
| Listing 16.3.3 | Inclusion/Exclusion and Eligibility | Listing of Subject Eligibility All Subjects Enrolled) |
| Listing 16.4 | Demographic Parameters | Listing of Demographic Parameters (All Subjects Enrolled) |
| Listing 16.5 | Routine Pre-procedure Testing Data | Listing of Routine Pre-procedure Testing Data (All Subjects Enrolled) |
| Listing 16.6 | Subject Evaluation Parameters | Listing of Subject Evaluation Parameters (All Subjects Enrolled) |
| Listing 16.7 | Subject Laboratory Parameters | Listing of Subject Laboratory Analysis Parameters (All Subjects Enrolled) |
| Listing 16.8 | Concomitant Medications | Listing of Concomitant Medications (All Subjects Enrolled) |
| Listing 16.9 | Procedure Evaluation | Listing of Procedure Evaluation Parameters (All Subjects Enrolled) |
| Listing 16.10.1 | Adverse Events During the Procedure | Listing of Adverse Events during Procedure (All Subjects Enrolled) |
| Listing 16.10.2 | MedDRA coding During the Procedure | Listing of MedDRA coding AE during Procedure (All Subjects Enrolled) |
| Listing 16.11 | Adverse Events Post-procedure Assessment | Listing of Adverse Events Post-procedure Assessment (All Subjects Enrolled) |
| Listing 16.12.1 | Adverse Events Post-procedure | Listing of Adverse Events Post-procedure (All Subjects Enrolled) |
| Listing 16.12.2 | MedDRA coding Post Procedure | Listing of MedDRA coded Adverse Events Post-Procedure (All Subjects Enrolled) |
| Listing 16.13.1 | Procedure Parameters-Pre-procedure | Listing of Input Parameters Pre-procedure (All Subjects Enrolled) |
| Listing 16.13.2 | Procedure Parameters-Pre-procedure | Listing of Estimator Parameters Pre-procedure (All Subjects Enrolled) |
| Listing 16.13.3 | Input Parameter | Listing of Input Procedure Parameters (All Subjects Enrolled) |
| Listing 16.14 | Procedure Parameters-End of Depletion Phase | Listing of End of Depletion Phase Parameters (All Subjects Enrolled) |
| Listing 16.15.1 | Procedure Results | Listing of Procedure Results (All Subjects Enrolled) |
| Listing 16.15.2 | Procedure Results | Listing of Procedure Results (All Subjects Enrolled) |
| Listing 16.16 | Primary Endpoint | Listing of Primary Endpoint (All Subjects Enrolled) |
| Listing 16.17.1 | Secondary Endpoint | Listing of Secondary Endpoints (All Subjects Enrolled) |
| Listing 16.17.2 | Secondary Endpoint | Listing of Waste Material for Secondary Endpoints (All Subjects Enrolled) |
| Listing 16.17.3 | End Hematocrit | Listing of End Hematocrit (All Subject Enrolled) |
| Listing 16.18 | Replacement RBC Unit Parameters | Listing of Replacement RBC Unit Parameters (All Subject Enrolled |

<sup>&</sup>lt;sup>1</sup>Titles for pediatric and adult subjects should be used for populating their respective output.

<sup>&</sup>lt;sup>2</sup>Summary of Empirical RBC Mass Balance Excluding Outlier(s) Table is provided for overall population only.

| Listing Number | Section | Description of Output |
|---|---|---|
| Listing 16.19 | Device Alarms | Listing of Device Alarms (All Subjects Enrolled) |
| Listing 16.20 | Waste Material-RBC Depletion/Exchange | Listing of Waste Material-RBC Depletion/Exchange Procedures (All Subjects Enrolled) |
| Listing 16.21 | Waste Material-RBC Exchange | Listing of Waste Material-RBC Exchange (All Subjects Enrolled) |
| Listing 16.22 | Protocol Deviations | Listing of Protocol Deviation (All Subjects Enrolled) |

## 10 MOCK TABLES AND LISTINGS

Table 14.1 Summary of Subject Disposition All Subjects Enrolled (N=xx)

| Parameter | Overall |
|----------------------------------|---------|
| Total Subjects | XX |
| Lead-In Subjects | XX |
| Intent-to-Treat Subjects | XX |
| Evaluable Subjects | XX |
| RBC Exchange Procedure | XX |
| RBC Depletion/Exchange Procedure | XX |
| Non-Evaluable Subjects | XX |
| RBC Exchange Procedure | XX |
| RBC Depletion/Exchange Procedure | XX |

Clinical Study Protocol: AMIC-003-CMD

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done

Table Status: DRAFT; SAS Program: Table 14.1.sas

Cross reference: Listing 16.1

Version: 21 Feb 2018

Table 14.2.1 Summary of Procedure Evaluability Intent-to-Treat Subjects<sup>1</sup> (N=xx)

| | Overall |
|---|---|
| | n (%) |
| Was the procedure completed? | |
| Yes | xx (%) |
| No | xx (%) |
| If No, check the primary reason: | |
| Adverse Event | xx (%) |
| Venous Access Issue (Non-Adverse Event) | xx (%) |
| Instrument Alarm | xx (%) |
| Disposable Issue | xx (%) |
| Leak | xx (%) |
| Kink | xx (%) |
| Misassembly | xx (%) |
| Other | xx (%) |
| Investigator Decision | xx (%) |
| Subject Decision | xx (%) |
| Protocol Deviation/Violation | xx (%) |
| Other | xx (%) |
| At the end of procedure, was reinfusion performed? | |
| Yes | xx (%) |
| No | xx (%) |
| NA | xx (%) |
| If Yes, was the subject's post-procedure blood sample taken prior to reinfusion? | |
| Yes | xx (%) |
| No | xx (%) |
| Did operator change subject Hct, Avg RF Hct, or Total Blood Volume after procedure start? | |
| Yes | xx (%) |
| No | xx (%) |
| NA | xx (%) |
| Was saline bolus performed? <sup>2</sup> | |
| Yes | xx (%) |
| No | xx (%) |
| NA | xx (%) |
| Is absolute difference of Average RF Hct and calculated Avg RF Hct≤5 Hct points? | |
| Yes | xx (%) |
| No | xx (%) |
| NA | xx (%) |
| Is absolute difference of subject Hct and pre-procedure Hct value ≤ 5 Hct points? | |
| Yes | xx (%) |
| No | xx (%) |
| NA | xx (%) |
| Is absolute difference of the FCR and calculated FCR value ≤ 6 FCR points? <sup>3</sup> | |
| Yes | xx (%) |
| No | xx (%) |
| NA | xx (%) |

Clinical Study Protocol: AMIC-003-CMD

Intent-to-Treat population is all subjects enrolled minus Lead-In subjects.

If a saline bolus is given during the procedure, the end Hct is not evaluable.

If Fraction of Cells Remaining was not used as an input, the evaluability criterion is not applicable.

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.2.1sas Cross reference: Listing 16.2 and 16.13.3

Table 14.2.2 Summary of Procedure Selection Parameters All Subjects Enrolled (N=xx)

| | | Overall<br>n (%) |
|--------------|---------------------------------|------------------|
| Is this a Lo | ead-In procedure? | |
| | Yes | xx (%) |
| | No | xx (%) |
| If Yes | | |
| | Lead-in RBC Exchange | xx (%) |
| | Lead-in RBC Depletion /Exchange | xx (%) |
| If No | | |
| | RBC Exchange | xx (%) |
| | RBC Depletion/ Exchange | xx (%) |

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.2.2sas

Cross reference: Listing 16.1

Table 14.3 Summary of Demographic Parameters All Subjects Enrolled (N=xx)

| Parameter | Overall |
|-------------------------------------------|--------------|
| Age at Consent (years) | |
| N | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| Min, Max | XX, XX |
| Age at Procedure (years) <sup>1</sup> | |
| N | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| Min, Max | XX, XX |
| Sex [n (%)] | |
| Male | xx (%) |
| Female | xx (%) |
| Ethnicity [n (%)] | |
| Hispanic or Latino | xx (%) |
| Not Hispanic or Latino | xx (%) |
| Decline to Respond | xx (%) |
| Race [n (%)] | |
| American Indian or Alaska Native | xx (%) |
| Asian | XX (%) |
| Black or African American | XX (%) |
| Native Hawaiian or Other Pacific Islander | XX (%) |
| White | XX (%) |
| Decline to Respond | xx (%) |

<sup>1</sup> For calculated parameters refer to algorithm document (AD) Note: NA=Not Applicable; UNK=Unknown; ND=Not Done

Table Status: DRAFT; SAS Program: Table 14.3.sas

Cross reference: Listing 16.4

Table 14.4
Summary of Routine Pre-Procedure Testing Data
Intent-to-Treat Subjects (N=xx)

| Parameter | N | Mean (SD) | Median | Min, Max |
|--------------------------------------|----|--------------|--------|----------|
| Actual Hemoglobin S (%) | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Target Hemoglobin S (%) <sup>1</sup> | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Hematocrit (%) | XX | xx.x (xx.xx) | XX.XX | XX, XX |

<sup>1</sup>Operator may input either Replacement Volume or FCR. For those that enter by Replacement Volume, a Target HbS value is not necessary

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.4.sas

Cross reference: Listing 16.5

Table 14.5 Summary of Subject Evaluations Parameters All Subjects Enrolled (N=xx)

| Parameter | N | Mean (SD) | Median | Min, Max |
|---|---|---|---|---|
| Weight (lb) | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Height (in) | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Systolic Blood Pressure (mmHg) | | | | |
| Pre-Procedure | xx | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| End of Depletion Phase <sup>1</sup> | XX | xx.xx (xx.xxx) | XX.XX | xx.x, xx.x |
| Post-Procedure | XX | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Diastolic Blood Pressure (mmHg) | | | | |
| Pre-Procedure | xx | xx.xx (xx.xxx) | XX.XX | xx.x, xx.x |
| End of Depletion Phase <sup>1</sup> | XX | xx.xx (xx.xxx) | xx.xx | xx.x, xx.x |
| Post-Procedure | XX | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Temperature (°F) | | | | |
| Pre-Procedure | XX | xx.xx (xx.xxx) | xx.xx | xx.x, xx.x |
| End of Depletion Phase <sup>1</sup> | XX | xx.xx (xx.xxx) | xx.xx | xx.x, xx.x |
| Post-Procedure | XX | xx.xx (xx.xxx) | XX.XX | xx.x, xx.x |
| Pulse (bpm) | | | | |
| Pre-Procedure | XX | xx.xx (xx.xxx) | xx.xx | xx.x, xx.x |
| End of Depletion Phase <sup>1</sup> | xx | xx.xx (xx.xxx) | xx.xx | xx.x, xx.x |
| Post-Procedure | xx | xx.xx (xx.xxx) | XX.XX | xx.x, xx.x |
| Respiration Rate (breaths/min) | | | | |
| Pre-Procedure | xx | xx.xx (xx.xxx) | xx.xx | xx.x, xx.x |
| End of Depletion Phase <sup>1</sup> | xx | xx.xx (xx.xxx) | xx.xx | xx.x, xx.x |
| Post-Procedure | XX | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |

<sup>1</sup>Additional analysis recorded at end of Depletion Phase for RBC Depletion/Exchange procedures

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done

Table Status: DRAFT; SAS Program: Table 14.5.sas

Cross reference: Listing 16.6

#### Table 14.6 Summary of Subject Laboratory Parameters All Subjects Enrolled (N=xx)

| Parameter | N | Mean (SD) | Median | Min, Max |
|---|---|---|---|---|
| White Blood Cell Count (WBC) (x10 <sup>3</sup> /μL) | | | | |
| Pre-Procedure | XX | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| End of Depletion Phase <sup>1</sup> | xx | xx.xx (xx.xxx) | XX.XX | xx.x, xx.x |
| Post-Procedure | xx | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Red Blood Cell Count (RBC) (x106/μL) | | | | |
| Pre-Procedure | XX | xx.xx (xx.xxx) | XX.XX | xx.x, xx.x |
| End of Depletion Phase <sup>1</sup> | XX | xx.xx (xx.xxx) | XX.XX | xx.x, xx.x |
| Post-Procedure | XX | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Platelet Count (x10 <sup>3</sup> /μL) | | | | |
| Pre-Procedure | XX | xx.xx (xx.xxx) | XX.XX | xx.x, xx.x |
| End of Depletion Phase <sup>1</sup> | XX | xx.xx (xx.xxx) | XX.XX | xx.x, xx.x |
| Post-Procedure | XX | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Hematocrit (%) | | | | |
| Pre-Procedure | XX | xx.xx (xx.xxx) | XX.XX | xx.x, xx.x |
| End of Depletion Phase <sup>1</sup> | xx | xx.xx (xx.xxx) | xx.xx | xx.x, xx.x |
| Post-Procedure | XX | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Plasma Hemoglobin (mg/dL) | | | | |
| Pre-Procedure | xx | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| End of Depletion Phase <sup>1</sup> | xx | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Post-Procedure | XX | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Hemoglobin A <sup>2</sup> (%) | | | | |
| Pre-Procedure | xx | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Post-Procedure | XX | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Hemoglobin S <sup>2</sup> (%) | | | | |
| Pre-Procedure | xx | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Post -Procedure | XX | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Hemoglobin C <sup>2</sup> (%) | | | | |
| Pre-Procedure | xx | xx.xx (xx.xxx) | xx.xx | xx.x, xx.x |
| Post -Procedure | XX | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Hemoglobin F <sup>2</sup> (%) | | | | |
| Pre-Procedure | xx | xx.xx (xx.xxx) | xx.xx | xx.x, xx.x |
| Post -Procedure | XX | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |
| Hemoglobin A2 <sup>2</sup> (%) | | | | |
| Pre-Procedure | xx | xx.xx (xx.xxx) | XX.XX | xx.x, xx.x |
| Post -Procedure | XX | xx.xx (xx.xxx) | XX.XX | XX.X, XX.X |

Clinical Study Protocol: AMIC-003-CMD

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done

Table Status: DRAFT; SAS Program: Table 14.6.sas

Cross reference: Listing 16.7

<sup>&</sup>lt;sup>1</sup>Additional analysis recorded at end of Depletion Phase for RBC Depletion/Exchange procedures

<sup>&</sup>lt;sup>2</sup>Only Hemoglobin values that could be quantified were entered into the database.

Table 14.7 Analysis of Primary Endpoint Parameters All Evaluable Subjects (N=xx)

| Parameter | N | Mean (SD) | Median | Min,Max | 95% CI |
|---|---|---|---|---|---|
| Post-Procedure Hemoglobin S (%) | XX | xx.x (xx.xx) | XX.XX | xx, xx | |
| Pre-Procedure Hemoglobin S (%) | xx | xx.x (xx.xx) | XX.XX | xx, xx | |
| Actual FCR <sup>1</sup> (%) | xx | xx.x (xx.xx) | XX.XX | xx, xx | |
| FCR (%) | XX | xx.x (xx.xx) | XX.XX | xx, xx | |
| Calculated A:T FCR Ratio <sup>1</sup> | xx | xx.x (xx.xx) | XX.XX | xx, xx | x.xx, x.xx |

<sup>1</sup>For calculated parameters refer to the algorithm document (AD) Note: NA=Not Applicable; UNK=Unknown; ND=Not Done

Table Status: DRAFT; SAS Program: Table 14.7.sas

Cross reference: Listing 16.16

Table 14.8
Summary of Secondary Endpoint Parameters
All Evaluable Subjects (N=xx)

| Parameter <sup>1</sup> | N | Mean (SD) | Median | Min,Max |
|---|---|---|---|---|
| Overall Procedures | | | | |
| Subject WBC Percent Loss <sup>2</sup> (%) | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Subject RBC Percent Loss <sup>2</sup> (%) | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Subject Platelet Percent Loss <sup>2</sup> (%) | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Subject Plasma Hemoglobin Delta (mg/dL) | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Calculated Target End Hct Accuracy (%) | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Exchange Procedures | | | | |
| Waste Material Volume (mL) | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Waste WBC Count (x10 <sup>10</sup> ) | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Waste Platelet Count (x10 <sup>11</sup> ) | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Calculated Target End Hct Accuracy (%) | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Depletion/Exchange Procedure | | | | |
| <b>Depletion Phase</b> | | | | |
| Waste Material Volume (mL) | xx | xx.x (xx.xx) | xx.xx | xx, xx |
| Waste WBC Count (x10 <sup>10</sup> ) | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Waste Platelet Count $(x10^{11})$ | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Calculated Depletion Hct Accuracy (%) | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Exchange Phase | | , , | | |
| Waste Material Volume (mL) | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Waste WBC Count (x10 <sup>10</sup> ) | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Waste Platelet Count (x10 <sup>11</sup> ) | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Calculated Target End Hct Accuracy (%) | XX | xx.x (xx.xx) | xx.xx | xx, xx |

<sup>1</sup>For calculated parameters refer to algorithm document (AD)

<sup>2</sup>For Subject Percent Loss, negative values indicate a gain

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done

Table Status: DRAFT; SAS Program: Table 14.8.sas

Cross reference: Listing 16.17.1 and 16.17.2

Table 14.9
Summary of Procedure Evaluation Parameters
All Evaluable Subjects (N=xx)

| Parameter | N | Mean (SD) | Median | Min, Max |
|---|---|---|---|---|
| Blood Warmer Prime Volume (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Subject Total Sample Volume Removed (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done

Table Status: DRAFT; SAS Program: Table 14.9.sas

Cross reference: Listing 16.9

Table 14.10.1
Summary of Adverse Events During the Procedure
All Subjects Enrolled (N=xx)

| Adverse Event Parameter | Subjects <sup>1</sup> | Events<br>n |
|---------------------------|-----------------------|-------------|
| Level | n (%) | |
| Total | xx (xx.x) | XX |
| Severity <sup>2</sup> | | |
| Mild | xx (xx.x) | XX |
| Moderate | xx (xx.x) | XX |
| Severe | xx (xx.x) | XX |
| Serious | | |
| Yes | xx (xx.x) | XX |
| No | xx (xx.x) | XX |
| Relationship to Procedure | | |
| Not Related | xx (xx.x) | XX |
| Unlikely Related | xx (xx.x) | XX |
| Possibly Related | xx (xx.x) | xx |
| Related | xx (xx.x) | xx |
| Relationship to Device | | |
| Not Related | xx (xx.x) | XX |
| Unlikely Related | xx (xx.x) | XX |
| Possibly Related | xx (xx.x) | XX |
| Related | xx (xx.x) | XX |

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.10.1.sas

Cross reference: Listing 16.10.1

<sup>&</sup>lt;sup>1</sup>Number of subjects experiencing one or more adverse events.

<sup>&</sup>lt;sup>2</sup>Subjects experiencing multiple events with different severity levels are counted only once for the most severe condition.
Table 14.10.2 Summary of Adverse Events During the Procedure by Site All Subjects Enrolled (N=xx)

| Site | Adverse Event Parameter<br>Level | Subjects <sup>1</sup> n (%) | Events<br>n |
|---|---|---|---|
| BCW (N=xx) | Total | xx (xx.x) | XX |
| | Severity <sup>2</sup> | | |
| | Mild | xx (xx.x) | xx |
| | Moderate | xx (xx.x) | xx |
| | Severe | xx (xx.x) | XX |
| | Serious | | |
| | Yes | xx (xx.x) | XX |
| | No | xx (xx.x) | XX |
| | Relationship to Procedure | | |
| | Not Related | xx (xx.x) | XX |
| | Unlikely Related | xx (xx.x) | XX |
| | Possibly Related | xx (xx.x) | XX |
| | Related | xx (xx.x) | XX |
| | Relationship to Device | | |
| | Not Related | xx (xx.x) | XX |
| | Unlikely Related | xx (xx.x) | XX |
| | Possibly Related | xx (xx.x) | XX |
| | Related | xx (xx.x) | XX |

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.10.2.sas

Cross reference: Listing 16.10.1

<sup>&</sup>lt;sup>1</sup>Number of subjects experiencing one or more adverse events.

<sup>&</sup>lt;sup>2</sup>Subjects experiencing multiple events with different severity levels are counted only once for the most severe condition.

## Table 14.10.3 Incidence of Adverse Events During the Procedure All Subjects Enrolled (N=xx)

| Adverse Events Reported <sup>1</sup> | | | |
|---|---|---|---|
| MedDRA | | | |
| System Organ Class Preferred Term Subjects <sup>2</sup> Events n (%) n | | | |
| Chills | Chills | xx (xx.x) | XX |
| Headache | Headache | xx (xx.x) | XX |
| Muscle Discomfort | Muscle Discomfort | xx (xx.x) | XX |
| Skin Irritation | Skin Irritation | xx (xx.x) | XX |
| Fainting | Fainting | xx (xx.x) | XX |

Clinical Study Protocol: AMIC-003-CMD

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.10.3.sas

Cross reference: Listing 16.10.2

<sup>&</sup>lt;sup>1</sup>Adverse events are sorted in descending frequency of events

<sup>&</sup>lt;sup>2</sup>Subjects experiencing multiple episodes of a given adverse event are counted only once for each adverse event term.

Table 14.10.4
Incidence of Adverse Events during the Procedure by Site
All Subjects Enrolled (N=xx)

| | Adverse Events Reported1 | | | |
|---|---|---|---|---|
| Site | MedDRA | | | |
| | System Organ Class | Preferred Term | Subjects <sup>2</sup><br>n (%) | Events<br>n |
| BCW<br>(N=xx) | Nervous system disorders | Dizziness | xx (xx.x) | XX |
| | Eye disorders | Vision blurred | xx (xx.x) | xx |
| | Gastrointestinal disorders | Nausea | xx (xx.x) | xx |
| | General disorders and administration site conditions | Chest pain | xx (xx.x) | xx |
| | Investigations | Blood pressure decreased | xx (xx.x) | XX |
| | Musculoskeletal and connective tissue disorders | Back pain | xx (xx.x) | xx |

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.10.4.sas

Cross reference: Listing 16.10.2

<sup>&</sup>lt;sup>1</sup> Adverse events are sorted in descending frequency of events

<sup>&</sup>lt;sup>2</sup>Subjects experiencing multiple episodes of a given adverse event are counted once for each adverse event term.

Table 14.11.1 Summary of Adverse Events Post-Procedure All Subjects Enrolled (N=xx)

| Adverse Event Parameter<br>Level | Subjects <sup>1</sup><br>n (%) | Events<br>n |
|---|---|---|
| Total | xx (xx.x) | xx |
| Severity <sup>2</sup> | | |
| Mild | xx (xx.x) | XX |
| Moderate | xx (xx.x) | XX |
| Severe | xx (xx.x) | XX |
| Serious | | |
| Yes | xx (xx.x) | XX |
| No | xx (xx.x) | XX |
| Relationship to Procedure | | |
| Not Related | xx (xx.x) | XX |
| Unlikely Related | xx (xx.x) | XX |
| Possibly Related | xx (xx.x) | XX |
| Related | xx (xx.x) | XX |
| Relationship to Device | | |
| Not Related | xx (xx.x) | XX |
| Unlikely Related | xx (xx.x) | XX |
| Possibly Related | xx (xx.x) | XX |
| Related | xx (xx.x) | XX |

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.11.1.sas

Cross reference: Listing 16.12.1

<sup>&</sup>lt;sup>1</sup>Number of subjects experiencing one or more adverse events.

<sup>&</sup>lt;sup>2</sup>Subjects experiencing multiple events with different severity levels are counted only once for the most severe condition

Table 14.11.2 Summary of Adverse Events Post-Procedure by Site All Subjects Enrolled (N=xx)

| Site | Adverse Event Parameter<br>Level | Subjects <sup>1</sup><br>n (%) | Events<br>n |
|---|---|---|---|
| BCW (N=xx) | Total | xx (xx.x) | XX |
| | Severity <sup>2</sup> | | |
| | Mild | xx (xx.x) | xx |
| | Moderate | xx (xx.x) | xx |
| | Severe | xx (xx.x) | xx |
| | Serious | | |
| | Yes | xx (xx.x) | xx |
| | No | xx (xx.x) | xx |
| | Relationship to Procedure | | |
| | Not Related | xx (xx.x) | xx |
| | Unlikely Related | xx (xx.x) | XX |
| | Possibly Related | xx (xx.x) | xx |
| | Related | xx (xx.x) | xx |
| | Relationship to Device | | |
| | Not Related | xx (xx.x) | xx |
| | Unlikely Related | xx (xx.x) | XX |
| = | Possibly Related | xx (xx.x) | XX |
| | Related | xx (xx.x) | XX |

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.11.2.sas

Cross reference: Listing 16.12.1

<sup>&</sup>lt;sup>1</sup>Number of subjects experiencing one or more adverse events.

<sup>&</sup>lt;sup>2</sup>Subjects experiencing multiple events with different severity levels are counted only once for the most severe condition.

#### Table 14.11.3 Incidence of Adverse Events Post-Procedure All Subjects Enrolled (N=xx)

| Adverse Events Reported <sup>1</sup> | | | |
|---|---|---|---|
| MedDRA | | | |
| System Organ Class Preferred Term Subjects <sup>2</sup> Events n (%) | | | |
| Chills | Chills | xx (xx.x) | XX |
| Headache | Headache | xx (xx.x) | XX |
| Muscle Discomfort | Muscle Discomfort | xx (xx.x) | XX |
| Skin Irritation | Skin Irritation | xx (xx.x) | XX |
| Fainting | Fainting | xx (xx.x) | XX |

Clinical Study Protocol: AMIC-003-CMD

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.11.3.sas

Cross reference: Listing 16.12.2

<sup>&</sup>lt;sup>1</sup>Adverse events are sorted in descending frequency of events.

<sup>&</sup>lt;sup>2</sup>Subjects experiencing multiple episodes of a given adverse event are counted once for each adverse event term.

#### Table 14.11.4 Incidence of Adverse Events Post-Procedure by Site All Subjects Enrolled (N=xx)

| | Adverse Events Reported <sup>1</sup> | | | |
|---|---|---|---|---|
| G:4 - | MedDRA | | | |
| Site | System Organ Class | Preferred Term | Subjects <sup>2</sup> n (%) | Events<br>n |
| BCW (N=xx) | Nervous system disorders | Dizziness | xx (xx.x) | XX |
| | Eye disorders | Vision blurred | xx (xx.x) | XX |
| | Gastrointestinal disorders | Nausea | xx (xx.x) | xx |
| | General disorders and administration site conditions | Chest pain | xx (xx.x) | XX |
| | Investigations | Blood pressure decreased | xx (xx.x) | XX |
| | Musculoskeletal and connective tissue disorders | Back pain | xx (xx.x) | XX |

Clinical Study Protocol: AMIC-003-CMD

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done

Table Status: DRAFT; SAS Program: Table 14.11.4.sas

Cross reference: Listing 16.12.2

<sup>&</sup>lt;sup>1</sup>Adverse events are sorted in descending frequency of events.

<sup>&</sup>lt;sup>2</sup>Subjects experiencing multiple episodes of a given adverse event are counted once for each adverse event term.

Table 14.12.1 Summary of Input and Estimator Parameters All Evaluable Subjects (N=xx)

| Parameter | N | Mean (SD) | Median | Min, Max |
|---|---|---|---|---|
| Input Pre-Procedure | | | | |
| FCR (%) | xx | xx.x (xx.xx) | XX.X | xx, xx |
| End Hematocrit (%) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Depletion Hematocrit (%) <sup>1</sup> | xx | xx.x (xx.xx) | XX.X | xx, xx |
| Replacement Volume (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Fluid Balance (mL) | xx | xx.x (xx.xx) | XX.X | xx, xx |
| AC Ratio | xx | xx.x (xx.xx) | XX.X | xx, xx |
| Start Prime Hematocrit (%) | xx | xx.x (xx.xx) | XX.X | xx, xx |
| End Prime Hematocrit (%) | xx | xx.x (xx.xx) | XX.X | XX, XX |
| Estimator | | | | |
| Whole Blood Flow Rate (mL/min) | xx | xx.x (xx.xx) | XX.X | xx, xx |
| Procedure Time (min) | xx | xx.x (xx.xx) | XX.X | xx, xx |
| Anticoagulant to Subject (mL) | xx | xx.x (xx.xx) | XX.X | xx, xx |
| Anticoagulant Used (mL) | xx | xx.x (xx.xx) | XX.X | xx, xx |
| Other Replacement Fluid (mL) <sup>1</sup> | xx | xx.x (xx.xx) | XX.X | xx, xx |
| Depletion Red Cell Volume (mL) <sup>1</sup> | XX | xx.x (xx.xx) | XX.X | XX, XX |
| Input | | | | |
| Subject Hematocrit (%) | xx | xx.x (xx.xx) | xx.x | xx, xx |
| Was value changed during procedure? | | | | |
| Yes | xx | | | |
| No | xx | | | |
| 2.0 | | | | |
| Total Blood Volume (mL) | xx | xx.x (xx.xx) | XX.X | XX, XX |
| Was value changed during procedure? | | | | |
| Yes | xx | | | |
| No | xx | | | |
| Maximum Whole Blood Flow Rate (mL/min) | XX | xx.x(xx.xx) | XX.X | XX, XX |
| Was value changed during procedure? | | | | |
| Yes | XX | | | |
| No | XX | | | |
| Citrate Infusion Rate (CIR) (mg/kg/min) | xx | xx.x (xx.xx) | xx.x | xx, xx |
| Was value changed during procedure? | 1878 | | | |
| Yes | xx | | | |
| No | XX | | | |
| Average Replacement Fluid Hematocrit (%) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Was value changed during procedure? | , AA | interior (interior) | | |
| Was value changed during procedure: Yes | XX | | | |
| No | XX | | | |

Clinical Study Protocol: AMIC-003-CMD

Parameter applies to RBC Depletion/Exchange procedures
Note: NA=Not Applicable; UNK=Unknown; ND=Not Done; AC=anticoagulant
Table Status: DRAFT; SAS Program: Table 14.12.1.sas
Cross reference: Listing 16.13.1, 16.13.2 and 16.13.3

Table 14.12.2
Summary of Procedure Parameters End of Depletion Phase<sup>1</sup>
All Evaluable Subjects (N=xx)

| Parameter | N | Mean (SD) | Median | Min, Max |
|---|---|---|---|---|
| Fluid Balance (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Depletion Hematocrit (%) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Whole Blood Processed (mL) | XX | xx.x (xx.xx) | XX.X | XX, XX |
| Replacement Fluid Albumin Returned (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Replacement Fluid Saline Returned (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Custom Replacement Fluid Returned (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Plasma Returned (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Procedure Time (minutes) | XX | xx.x (xx.xx) | XX.X | XX, XX |
| Anticoagulant Used (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Anticoagulant to Subject (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Saline to Subject (mL) | XX | xx.x (xx.xx) | XX.X | XX, XX |

<sup>1</sup>Applicable for RBC Depletion/Exchange procedures Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.12.2.sas

Cross reference: Listing 16.14

Table 14.13.1 Summary of Procedure Results All Evaluable Subjects (N=xx)

| Parameter | N | Mean (SD) | Median | Min, Max |
|---|---|---|---|---|
| Procedure Time (minutes) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| FCR (%) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| A:T FCR Ratio <sup>1</sup> | XX | xx.x (xx.xx) | XX.X | xx, xx |
| End Hematocrit (%) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Fluid Balance (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Theoretical RBC Mass Balance (mL) <sup>1</sup> | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Empirical RBC Mass Balance (mL) <sup>1</sup> | XX | xx.x (xx.xx) | xx.x | xx, xx |
| Whole Blood Processed (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Replacement Fluid to Subject (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Anticoagulant to Subject (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Anticoagulant Used (mL) | XX | xx.x (xx.xx) | XX.X | XX, XX |
| Saline to Subject (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Replacement Fluid Albumin Returned (mL) <sup>2</sup> | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Replacement Fluid RBC Returned (mL) | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Replacement Fluid Saline Returned (mL) <sup>2</sup> | XX | xx.x (xx.xx) | XX.X | xx, xx |
| Custom Replacement Fluid Returned (mL) <sup>2</sup> | XX | xx.x (xx.xx) | XX.X | xx, xx |

<sup>1</sup>For calculated parameters refer to algorithm document (AD)

<sup>2</sup>Applicable for RBC Depletion/Exchange Procedures

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done

Table Status: DRAFT; SAS Program: Table 14.13.1.sas

Cross reference: Listing 16.15.1 and 16.15.2

#### Table 14.13.2 Summary of Empirical RBC Mass Balance Excluding Outlier(s) All Evaluable Subjects (N=xx)

| Parameter | N | Mean (SD) | Median | Min, Max |
|---|---|---|---|---|
| Empirical RBC Mass Balance (mL) <sup>1,2</sup> | XX | xx.xxx (xxxx.xxxx) | XX.XXX | xx.xx,xx.xx |

Clinical Study Protocol: AMIC-003-CMD

<sup>1</sup>For calculated parameters refer to the algorithm document (AD)

<sup>2</sup>Excludes xx subjects with outlier values using Box and Whisker plot (Subject IDs xxxxx, ...)

Note: NA=Not Applicable: UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.13.2.sas

Cross reference: Listing 16.15.1 and 16.15.2

Table 14.14 Summary of Replacement RBC Unit Parameters All Evaluable Subjects (N=xx)

| Parameter | N | Mean (SD) | Median | Min, Max |
|---------------------------|----|--------------|--------|----------|
| Hematocrit (%) | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Volume (mL) <sup>1</sup> | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Plasma Hemoglobin (mg/dL) | XX | xx.x (xx.xx) | XX.XX | xx, xx |

<sup>1</sup>For calculated parameters refer to the algorithm document (AD) Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.14.sas

Cross reference: Listing 16.18

Table 14.15 Summary of Device Alarms All Subjects Enrolled (N=xx)

| Alarm | Frequency (Occurrence per Procedure) x | Total Number<br>of Procedures<br>n (%) |
|---|---|---|
| ACD Flow Problem | XX | xx (%) |
| Air Detected | XX | xx (%) |
| Blood Warmer Prime Flow Problem | XX | xx (%) |
| Cassette Pressure Limit Exceeded | XX | xx (%) |
| Centrifuge Line Blockage | XX | xx (%) |
| Check Replacement Fluids | XX | xx (%) |
| Empty ACD | XX | xx (%) |
| Return Line Occlusion | XX | xx (%) |
| Empty Saline | XX | xx (%) |
| Inlet Line Occlusion | XX | xx (%) |
| Other | xx | xx (%) |

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.15.sas

Cross reference: Listing 16.19

### Table 14.16.1 Summary of Waste Material-RBC Depletion/Exchanges All Evaluable Subjects (N=xx)

| | | RBC Deple | tion Phase | | | RBC Exch | ange Phase | • |
|---|---|---|---|---|---|---|---|---|
| Parameter | N | Mean (SD) | Median | Min,<br>Max | N | Mean (SD) | Median | Min,<br>Max |
| Volume (mL) <sup>1</sup> | XX | xx.x (xx.xx) | XX.XX | XX, XX | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| WBC $(x10^3/\mu L)$ | XX | xx.x (xx.xx) | XX.XX | XX, XX | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Total WBC Count (x10 <sup>10</sup> ) <sup>1</sup> | XX | xx.x (xx.xx) | XX.XX | XX, XX | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Platelet Count (x10 <sup>3</sup> /μL) | XX | xx.x (xx.xx) | xx.xx xx, xx | | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Total Platelet Count (x10 <sup>11</sup> ) <sup>1</sup> | XX | xx.x (xx.xx) | XX.XX | xx, xx | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Hematocrit (%) | XX | xx.x (xx.xx) | XX.XX | XX, XX | XX | xx.x (xx.xx) | XX.XX | XX, XX |

Clinical Study Protocol: AMIC-003-CMD

<sup>1</sup>For calculated parameters refer to the algorithm document (AD) Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.16.1.sas

Cross reference: Listing 16.20

Table 14.16.2 Summary of Waste Material - RBC Exchange Procedures All Evaluable Subjects (N=xx)

| Parameter | N | Mean (SD) | Median | Min, Max |
|---|---|---|---|---|
| Volume (mL) <sup>1</sup> | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| WBC $(x10^3/\mu L)$ | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Total WBC Count (x 10 <sup>10</sup> ) <sup>1</sup> | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Platelet Count (x10 <sup>3</sup> /μL) | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Total Platelet Count (x10 <sup>11</sup> ) <sup>1</sup> | XX | xx.x (xx.xx) | XX.XX | xx, xx |
| Hematocrit (%) | XX | xx.x (xx.xx) | XX.XX | xx, xx |

<sup>1</sup>For calculated parameters refer to the algorithm document (AD) Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Table Status: DRAFT; SAS Program: Table 14.16.2.sas

Cross reference: Listing 16.21

#### Table 14.17 Summary of End Hematocrit All Evaluable Subjects (N=xx)

| Parameter | N | Mean (SD) | Median | Min, Max |
|---|---|---|---|---|
| Target Depletion Hct (%) <sup>3</sup> | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Procedure Results Depletion Hct (%) <sup>1</sup> | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Subject Post-Depletion Phase Hct (%) <sup>2</sup> | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| End of Depletion Phase Hct Accuracy (%) <sup>5</sup> | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Target Exchange End Hct (%) <sup>3</sup> | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Procedure Results End Hct (%) <sup>4</sup> | XX | xx.x (xx.xx) | xx.xx | xx, xx |
| Subject Post-Procedure Hct (%) <sup>2</sup> | XX | xx.x (xx.xx) | xx.xx | XX, XX |
| End of Exchange Phase Hct Accuracy (%) 5 | XX | xx.x (xx.xx) | xx.xx | xx, xx |

Clinical Study Protocol: AMIC-003-CMD

Table Status: DRAFT; SAS Program: Table 14.17.sas

Cross reference: Listing 16.17.3

<sup>&</sup>lt;sup>1</sup>Depletion Hct (%) results reported Post-Depletion Phase

<sup>&</sup>lt;sup>2</sup>Subject laboratory measured values

<sup>&</sup>lt;sup>3</sup>Target Depletion Hct and Exchange End Hct values entered Pre-Procedure

<sup>&</sup>lt;sup>4</sup>End Hct (%) results reported Post-Procedure

<sup>&</sup>lt;sup>5</sup>For calculated parameters refer to algorithm document (AD) Note: NA=Not Applicable: UNK=Unknown; ND=Not Done

Listing 16.1 Listing of Patient Disposition All Subjects Enrolled (N=xx)

| | sts | | |
|---|---|---|---|
| Evaluable RBC | Depletion/Exchange Subject | Yes | |
| Evaluable RBC | <b>Exchange Subjects</b> | | No |
| Intent-to-Treat subjects <sup>1</sup> | | Yes | Lead-in |
| Subject | ID | XXXXX | XXXXX |

<sup>1</sup>Intent-to-Treat is defined as all subjects enrolled minus the Lead-In subjects. Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Listing Status: DRAFT; SAS Program: Listing 16.1.sas


Listing 16.2 Listing of Procedure Evaluability/End of Study All Subjects Enrolled (N=xx)

| | | | | | | | | Т | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Calculated<br>End Hct<br>Accuracy<br>Evaluable <sup>3</sup> | Evaluable | Non<br>Evaluable | Evaluable | Non<br>Evaluable | Evaluable | Evaluable | Evaluable | Evaluable | Evaluable | |
| Calculated<br>Depletion<br>Het<br>Accuracy<br>Evaluable <sup>3</sup> | Evaluable | Non<br>Evaluable | Evaluable | Non<br>Evaluable | Evaluable | Evaluable | Evaluable | Evaluable | Evaluable | |
| A:T FCR<br>Ratio<br>Evaluable <sup>3</sup> | Evaluable | Non<br>Evaluable | Evaluable | Non<br>Evaluable | Evaluable | Evaluable | Evaluable | Evaluable | Evaluable | |
| Is absolute difference of the FCR and calculated FCR value ≤ 6 FCR points?²⁴ | Yes | Yes | Yes | Yes | Yes | Yes | Yes | NA | No | |
| Is absolute difference of subject Hct and preprocedure Hct ≤ 5 Hct points?² | Yes | Yes | Yes | Yes | Yes | Yes | Yes | No | Yes | |
| Is absolute difference of Average RF Hct and calculated Avg RF Hct value ≤5 Hct points?2 | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | |
| Was<br>saline<br>bolus<br>perform<br>ed? <sup>1</sup> | No | No | No | No | Yes | No | No | No | No | |
| Did<br>operator<br>change<br>subject Hct,<br>Avg RF Hct,<br>or TBV<br>after<br>procedure<br>start? | No | No | No | Yes | No | No | No | No | No | |
| If Yes, was<br>the subject's<br>post-<br>procedure<br>blood sample<br>taken prior<br>to | NA | NA | No | NA | NA | NA | NA | NA | NA | |
| At the end<br>of the<br>procedure,<br>was<br>reinfusion<br>performed? | No | No | | | | | | | | - |
| If No,<br>reason<br>procedure<br>not<br>completed | NA | Adverse | NA | NA | NA | NA | NA | NA | NA | |
| Was<br>procedure<br>completed? | No | Yes | Yes | No | Yes | No | No | No | No | |
| Subject | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | |

If saline bolus is given during the procedure, the end Hct is not evaluable.

<sup>2</sup>For calculated parameters refer to algorithm document (AD)

<sup>3</sup>Lead-In subjects are not included in the evaluable population for this protocol

<sup>4</sup>If Fraction of Cells Remaining was not used as an input, the evaluability criterion is not applicable.

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done

FCR=fraction of cells remaining; Hb=hemoglobin; Hct=hematocrit; RF=replacement fluid

Listing Status: DRAFT; SAS Program: Listing 16.2.sas

Listing 16.3.1 Listing of Inclusion Criteria All Subjects Enrolled (N=xx)

| Subject<br>ID | Subject >6<br>years old | Subject Subject >6 Subject with SCD ID years old who require RBC Exchange or RBC Depletion/Exchange treatment | Medically stable<br>subjects treated for<br>SCD with RBC<br>Exchange or RBC<br>Depletion/Exchange | Subjects who have provided signed IC/assent prior to participation | Subjects who Adequate availability of sickle have provided trait negative, leukoreduced, signed IC/assent ABO blood group, Rh (D) rior to compatible, unexpired participation replacement RBC products | Subjects with sufficient vascular access for RBC procedure | Subjects with Subject is able and sufficient agrees to report AEs vascular access during the required for RBC reporting period procedure |
|---|---|---|---|---|---|---|---|
| XXXXX | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| XXXXX | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| XXXXX | No | No | No | No | No | No | No |
| XXXXX | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| | 74. J. D. 242.2 | CIVITY OUT THE TOTAL OF THE TOT | | | | | |

Clinical Study Protocol: AMIC-003-CMD
Note: NA=Not Applicable; UNK=Unknown; ND=Not Done
IC=informed consent; RBC=red blood cell; SCD=sickle cell disease
Listing Status: DRAFT; SAS Program: Listing 16.3.1.sas


Listing 16.3.2 Listing of Exclusion Criteria All Subjects Enrolled (N=xx)

| Subjects who fail to comply with site requirements for cessation of medication that interfere or increase procedure risk | No | No | No | No |
|---|---|---|---|---|
| Subjects<br>who are<br>pregnant | No | No | No | No |
| Subjects<br>who refuse<br>blood<br>products | No | No | No | No |
| Subjects who have a life expectanc y < 30 days | No | No | No | No |
| Subjects who had an SAE associated with an RBCx procedure in the past | No | No | No | No |
| Drug/alcohol abuse or other factors that could affect the ability of subject to comply with protocol requirements | No | No | No | No |
| Subjects with AMS that prohibit giving IC and assent and do not have LAR | No | No | No | No |
| Procedures<br>prescribed<br>within 1 wk<br>of hospital<br>discharge | No | No | No | No |
| Subject Procedures ID that occur during acute hospitaliza tion | No | No | No | No |
| Subject<br>ID | XXXXX | XXXXX | XXXXX | XXXXX |

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done

AMS=altered mental status; IC=informed consent; LAR=legally authorized representative; SAE=serious adverse event; wk=week Listing Status: DRAFT; SAS Program: Listing 16.3.2.sas


Listing 16.3.3 Listing of Subject Eligibility All Subjects Enrolled (N=xx)

| Subject ID | Has the subject met all eligibility criteria according to the protocol? | Date Informed Consent Signed |
|---|---|---|
| XXXXX | Yes, subject has met all eligibility criteria | Mmm-dd-yyyy |
| XXXXX | No, subject has not met all eligibility criteria | Mmm-dd-yyyy |
| XXXXX | Yes, subject has met all eligibility criteria | Mmm-dd-yyyy |
| XXXXX | No, subject has not met all eligibility criteria | Mmm-dd-yyyy |

Clinical Study Protocol: AMIC-003-CMD
Note: NA=Not Applicable; UNK=Unknown; ND=Not Done
Listing Status: DRAFT; SAS Program: Listing 16.3.3.sas


Listing of Demographic Parameters All Subjects Enrolled (N=xx) Listing 16.4

| Subject<br>ID | Date of<br>Birth | Age at<br>Consent<br>(years) | Age at Procedure (years) <sup>1</sup> | Sex | Ethnicity | Race |
|---|---|---|---|---|---|---|
| XXXXX | Mmm-dd-<br>yyyy | XX | xx | Male | Hispanic or<br>Latino | White |
| XXXXX | Mmm-dd-<br>yyyy | xx | XX | Female | Not Hispanic or<br>Latino | Black or African<br>American |
| XXXXX | Mmm-dd- | xx | xx | Female | Hispanic or<br>Latino | Asian |
| XXXXX | Mmm-dd- | XX | xx | Male | Hispanic or<br>Latino | Asian |
| XXXXX | Mmm-dd-<br>yyyy | XX | XX | Female | Not Hispanic or<br>Latino | American Indian<br>or Alaska Native |
| XXXXX | Mmm-dd- | XX | xx | Female | Hispanic or<br>Latino | Asian |
| XXXXX | Mmm-dd- | xx | xx | Male | Hispanic or<br>Latino | Decline to<br>Respond |
| XXXXX | Mmm-dd- | XX | xx | Female | Not Hispanic or<br>Latino | White |
| XXXXX | Mmm-dd- | XX | xx | Female | Hispanic or<br>Latino | Black or African<br>American |

Clinical Study Protocol: AMIC-003-CMD

For calculated parameters refer to algorithm document (AD)

Note: NA= Not Applicable; UNK= Unknown; ND= Not Done
Listing Status: DRAFT; SAS Program: Listing 16.4.sas


Listing of Routine Pre-Procedure Testing Data All Subjects Enrolled (N=xx)

| Γ | | | | | | | _ |
|---|---|---|---|---|---|---|---|
| | Hct (%) | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Target Hb S1 (%) | | XX.X | XXX.X | XX.X | XXX.X | XXX.X |
| | Actual Hb S (%) | | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Sample Time | (24 hour clock) | hh:mm | hh:mm | hh:mm | hh:mm | hh:mm |
| | Sample Date | | Mmm-dd-yyyy | Mmm-dd-yyyy | Mmm-dd-yyyy | Mmm-dd-yyyy | Mmm-dd-yyyy |
| | Subject ID | | XXXX | XXXX | XXXX | XXXX | XXXX |

Operator may input either Replacement Volume or FCR. For those that enter by Replacement Volume, a Target HbS value is not necessary. Note: NA=Not Applicable; UNK=Unknown; ND=Not Done; Hb=hemoglobin; Hct=hematocrit Listing Status: DRAFT; SAS Program: Listing 16.5.sas


Listing of Subject Evaluations Parameters All Subjects Enrolled (N=xx) Listing 16.6

| Subject<br>ID | Primary<br>Diagnosis | Procedure <sup>1</sup> | Weight (Ib) | Height (in) | Systolic BP<br>(mmHg) | Diastolic BP (mmHg) | Temp<br>(°F) | Pulse<br>(bpm) | Respiration<br>Rate<br>(breaths/min) |
|---|---|---|---|---|---|---|---|---|---|
| XXXXX | SS | Pre | XXX | XX | XXX | XXX | XX.X | XX | XXX |
| | | End of Depletion Phase | | | XXX | XXX | XX.X | XX | XXX |
| | | Post | | | XXX | XXX | XX.X | XX | XXX |
| XXXXX | SB-0 thal | Pre | XXX | XX | XXX | XXX | XX.X | XX | XXX |
| | | End of Depletion Phase | XXX | XXX | XXX | XXX | XXX.X | XXX | XXX |
| | | Post | XXX | XX | XXX | XXX | XX.X | XX | XXX |
| XXXXX | SC | Pre | XXX | XX | XXX | XXX | XX.X | XX | XXX |
| | | End of Depletion Phase | XXX | XX | XXX | XXX | XXX.X | X | XXX |
| | | Post | xxx | XX | XXX | XXX | XX.X | XX | XXX |
| XXXXX | Other | Pre | XXX | XX | XXX | XXX | XX.X | X | XXX |
| | | End of Depletion Phase | XXX | XX | XXX | XXX | xx.x | XX | XXX |
| | | Post | XXX | XX | XXX | XXX | XX.X | XX | XXX |
| XXXXX | SS | Pre | XXX | XX | XXX | XXX | XX.X | XX | XXX |
| | | End of Depletion Phase | XXX | XX | XXX | XXX | x.xx | XX | XXX |
| | | Post | XXX | XX | XXX | XXX | XX.X | XX | XXX |
| XXXXX | SS | Pre | XXX | XX | XXX | XXX | xx.x | XX | XXX |
| | | End of Depletion Phase | XXX | XX | xxx | xxx | XX.X | XX | XXX |
| | | Post | XXX | XX | XXX | XXX | XX.X | XX | XXX |
| Clinical Stu | dy Protocol. A | Tinical Study Protocol: AMIC-003-CMD | | | | | | | |

<sup>1</sup>Additional analysis recorded at end of Depletion Phase for RBC Depletion/Exchange procedures

Note: NA= Not Ápplicable; UNK= Unknown; ND= Not Done
BP=blood pressure; SB-0 thal= sickle beta 0 thalassemia; SC=sickle hemoglobin C disease; SS=sickle cell anemia; Temp=temperature
Listing Status: DRAFT; SAS Program: Listing 16.6.sas

Listing 16.7
Listing of Subject Laboratory Analysis Parameters
All Subjects Enrolled (N=xx)

| 2 | | T | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Pregnanc<br>y Test | Neg | | Q. | | Pos | | | | Male,<br>N/A | | QN | | Pos | | | | | |
| Post-<br>Procedu<br>re<br>Sample<br>Time <sup>3</sup> | | hh:mm | | hh:mm | | | | hh:mm | | hh:mm | | hh:mm | | | | : | hh:mm | |
| Hb A2 <sup>4</sup> (%) | XX.X | XX.X | XX.X | XX.X | XX.X | | | XX.X | XX.X | XX.X | XXX.X | XX.X | XX.X | | | | XX.X | |
| Hb F <sup>4</sup> (%) | XX.X | XX.X | XX.X | XX.X | XX.X | | | XX.X | XX.X | XX.X | X.XX | XX.X | X.X.X | | | | XX.X | |
| Hb C <sup>4</sup> (%) | XX.X | XX.X | XX.X | XX.X | XX.X | | | XX.X | XX.X | XX.X | X.XX | XX.X | XX.X | | | | XX.X | |
| Actual<br>FCR <sup>2</sup><br>(%) | | XX.X | | XX.X | | | | XX.X | | XX.X | | XX.X | | | | | XX.X | |
| Hb S <sup>4</sup> (%) | XX.X | XX.X | XX.X | XX.X | x.xx | | | XX.X | XX.X | XXX. | XXX.X | XX.X | XX.X | | | | XX.X | |
| Hb A⁴<br>(%) | XX.X | XX.X | XX.X | XX.X | XX.X | | | XXX.X | XXX.X | XX.X | XX | XX | xx | | | | XX | |
| Post-<br>Procedure<br>Sample Time <sup>3</sup> | | hh:mm | | hh:mm | | | | hh:mm | | hh:mm | | hh:mm | | | | | hh:mm | |
| Plasma<br>Hb<br>(mg/dL) | XX.X | XX.X | XX.X | XX.X | X.XX | XX.X | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | | | XX.X | |
| Post-<br>Procedure<br>Sample<br>Time <sup>3</sup> | | hh:mm | | hh:mm | | | | hh:mm | | hh:mm | | hh:mm | | | | | hh:mm | |
| Het<br>(%) | XX | X | xx | xx | XX | XX | | XX | XX | × | XX | XX | XX | xx | | | XX | |
| Platelet<br>Count<br>(x10³/µL) | XXX | XXX | XXX | XXX | xxx | XXX | | XXX | XXX | XXX | xxx | XXX | XXX | | | | XXX | |
| RBC (x106/µL) | xxx | XXX | XXX | XXX | XXX | XXX | | XXX | XXX | XXX | XXX | XXX | XXX | XXX | | | XXX | CAMD |
| WBC (x10³/µL) | xxx | XXX | XXX | XXX | XXX | XXX | | XXX | XXX | XXX | XXX | XXX | XXX | XXX | | | XXX | 1. ANATO OO |
| Procedure <sup>1</sup> | Pre | Post | Pre | Post | Pre | End of | Depletion<br>Phase | Post | Pre | Post | Pre | Post | Pre | End of | Depletion | Phase | Post | Citizani Str. dr. Dustonal, AMIC 002 CMD |
| Subje<br>ct<br>ID | XXXX | × | XXXX | × | XXXX | × | | | XXXX | < | XXXX | × | XXXX | | | | | 12 |

Clinical Study Protocol: AMIC-003-CMD <sup>1</sup>Additional analysis recorded at end of Depletion Phase for RBC Depletion/Exchange procedures

<sup>2</sup>For calculated parameters refer to algorithm document (AD)

<sup>3</sup>Sample time is 24 Hour clock

<sup>4</sup>Only Hemoglobin values that could be quantified were entered into the database.

Note: NA= Not Applicable; UNK= Unknown; ND= Not Done
FCR=fraction of cells remaining; Hb=hemoglobin; Hct=hematocrit; Neg=negative; Pos=positive; RBC=red blood cell; WBC=white blood cell
Listing Status: DRAFT; SAS Program: Listing 16.7.sas


# CONFIDENTIAL

Listing of Concomitant Medications All Subjects Enrolled (N=xx) Listing 16.8

| Subject | Any Con | Medication | Medication | Drug Class | Start | Continuing | End Date | Dose/ | Route | Frequency | Indication |
|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>a</b> | 110 | Verbatim <sup>2</sup> | (WHO Term) <sup>3</sup> | | Date | | | Unit | | | |
| XXXXX | Yes | Ca Gluconate CALCIUM | CALCIUM | CALCIUM | Mmm- | Yes | Mmm-dd- | | Topical | Morning | |
| | | | | GLUCONATE | dd-yyyy | | yyyy | | | | |
| XXXXX | Yes | Albuterol | | | Mmm- | No | Mmm-dd- | | Inhaled | As Needed | Asthma |
| | | | | | dd-yyyy | | уууу | | | | |
| | Yes | Benadryl | Benadryl | | Mmm- | No | Mmm-dd- | | IV | Other | |
| | | | | | dd-yyyy | | yyyy | | | | |

<sup>1</sup>Concomitant medications were not recorded for enrolled subjects that did not start a procedure.

<sup>2</sup>Medication is reported verbatim from the CRF.

<sup>3</sup>The medical terms are from WHO Drug Dictionary (version 2015).

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done
Listing Status: DRAFT; SAS Program: Listing 16.8.sas

Listing of Procedure Evaluation Parameters All Subjects Enrolled (N=xx) Listing 16.9

| Was procedure<br>ended prior to<br>or extended<br>beyond<br>(±50mLs) of the<br>Target RF | Yes | No | Yes | Yes |
|---|---|---|---|---|
| If Yes,<br>provide<br>the<br>prime<br>volume<br>(mL) | Yes | No | Yes | Yes |
| Was a blood warme r used during proced ure? | XX | XX | XX | xx |
| Was<br>prime<br>diverted<br>? | Yes | Yes | No | No |
| CP³ | Full | Partial | Full | None |
| STSVR (mL) | XX | XX | XX | XX |
| Was<br>reinfusion<br>selected<br>prior to<br>start of<br>procedure? | Yes | Yes | No | Yes |
| AC<br>Type | ACD- | Custo | Custo | ACD- |
| RF<br>Used <sup>2</sup> | Saline | Albumi | Saline | Custom |
| Venous<br>Access<br>Used | Central | hh:mm Peripher al | Central<br>and<br>Peripher<br>al | Central |
| End<br>Time <sup>1</sup> | hh:mm | hh:mm | hh:mm | hh:mm |
| Procedure<br>Date | Mmm-dd- | Mmm-dd-<br>yyyy | _ | Mmm-dd-<br>yyyy |
| Subject | XXXXX | XXXXX | XXXXX | XXXXX |

<sup>1</sup>End time is 24 Hour clock

<sup>2</sup> Applicable for Depletion/Exchange procedures

<sup>3</sup>Applicable for Exchange procedures
Note: NA= Not Applicable; UNK= Unknown; ND= Not Done
AC=anticoagulant; ACD-A=Anticoagulant Citrate Dextrose Formula A; CP= Custom Prime; RF=Replacement Fluid; STSVR=Subject Total Sample Volume

Removed

Listing Status: DRAFT; SAS Program: Listing 16.9.sas

Listing 16.10.1
Listing of Adverse Events During Procedure
All Subjects Enrolled (N=xx)

| Outco<br>me/<br>End<br>Date | Recove red/<br>Mmm-<br>dd-<br>yyyy | Contin | Contin | Recove red/<br>Mmm-<br>dd- | Contin |
|---|---|---|---|---|---|
| Serious<br>/Reaso<br>n | No | No | Yes/<br>Hospita<br>lization | No | Yes/<br>Death |
| Relationsh<br>ip to<br>Device | Not<br>Related | Not<br>Related | Possibly<br>Related | | Related |
| Relatio<br>nship<br>to<br>Proced<br>ure | Possibl<br>y<br>Related | Possibl<br>y<br>Related | Not<br>Related | Related | Unlikel<br>y<br>Related |
| Action<br>Taken<br>(Subject) | No | No | Yes | No | Yes |
| Action<br>Taken<br>(Procedure) | No Change | No Change | Interrupted | Change in<br>Parameters/<br>specify | Interrupted |
| Episode<br>Pattern | Single | Single | Cont | Single | Cont |
| Severity | Mild | Mild | Severe | Mild | Severe |
| Start<br>Date | Mmm-<br>dd-yyyy | Mmm-<br>dd-yyyy | Mmm-<br>dd-yyyy | Mmm-<br>dd-yyyy | Mmm-<br>dd-yyyy |
| Description<br>of Event | Nausea | Chills | Chills | Other:<br>specify | Chills |
| AE<br>Number | | | | | |
| Any<br>AEs? | Yes | Yes | Yes | Yes | Yes |
| Study<br>Site | BCW | BCW | NCH | UT | KCI |
| Subject<br>ID | XXXXX | XXXXX | XXXXX | XXXX | XXXXX |

Clinical Study Protocol: AMIC-003-CMD
Note: NA=Not Applicable; UNK=Unknown; ND=Not Done
AEs=adverse event
Listing Status: DRAFT; SAS Program: Listing 16.10.1.sas


Listing of MedDRA Coded Adverse Events During Procedure All Subjects Enrolled (N=xx)

| Sudy Site Adverse Event Event Mumber Description of Event Event Event Mumber System Organ Class Preferred Term Term Term Term High Level Low Level Term Term xxxxxx BCW Nausea Chills Chills Chills Chills xxxxxx BCW Chills Chills Chills Chills Chills | | | | | | MedDR | MedDRA Term | |
|---|---|---|---|---|---|---|---|---|
| BCW<br>BCW | Subject<br>ID | Study Site | Adverse<br>Event<br>Number | Description of<br>Event | System<br>Organ Class | Preferred<br>Term | High Level<br>Term | Low Level<br>Term |
| BCW BCW | XXXXX | BCW | | Nausea | | | | |
| BCW | XXXXX | BCW | | Chills | | | | |
| | XXXXX | BCW | | Other: specify | | | | |
| | XXXXX | | | Chills | | | | |

Clinical Study Protocol: AMIC-003-CMD
Note: NA=Not Applicable; UNK=Unknown; ND=Not Done
Listing Status: DRAFT; SAS Program: Listing 16.10.2.sas


 $\label{eq:control} Listing~16.11$  Listing of Adverse Events Post-Procedure Assessment All Subjects Enrolled (N=xx)

| experienc e any AE post- procedur e? | Yes | Yes | No |
|---|---|---|---|
| Death<br>(Date of<br>Death) | Mmm-dd-<br>yyyy | Mmm-dd-<br>yyyy | Mmm-dd-<br>yyyy |
| Continu | Yes | No | No |
| Recovered<br>with<br>Sequela(e)<br>(End Date) | Mmm-dd-<br>yyyy | Mmm-dd-<br>yyyy | Mmm-dd-<br>yyyy |
| Recover<br>ed (End<br>Date) | Mmm-<br>dd-yyyy | Mmm-<br>dd-yyyy | Mmm-<br>dd-yyyy |
| procedure with Outcome of Continuing? | Yes | No | No |
| by telephone, was a certified letter sent to the subject? | No. | Yes | Yes |
| time<br>of 2nd<br>contac<br>t <sup>1,2</sup> | Mmm-<br>dd-<br>yyyy<br>hh:mm | Mmm-<br>dd-<br>yyyy<br>hh:mm | Mmm-<br>dd-<br>yyyy<br>hh:mm |
| contacte<br>d on 2nd<br>attempt<br>? | N <sub>o</sub> | No | Yes |
| time of<br>1st<br>contact <sup>1</sup> , | Mmm-<br>dd-yyyy<br>hh:mm | Mmm-<br>dd-yyyy<br>hh:mm | Mmm-<br>dd-yyyy<br>hh:mm |
| contacted<br>on 1st<br>attempt? | Yes | Yes | No |
| | 00 | 15 | 16 |
| | XXXXX | XXXXX | XXXXX |
| | time of contacte time contacted procedure 1st don 2nd of 2nd by with ed (End Mith contact), attempt contact telephone, 2 | contacted time of contact time of contacted time of contacted time of contacted time of contact time of contact time of contact. Ist don 2nd of 2nd by with on 1st attempt? attempt? contact. attempt contact. at | contacted time of contacte time contacted procedure by with on 1st 1st don 2nd of 2nd by with on 1st 1st don 2nd of 2nd ed by with on 1st 1st don 2nd of 2nd ed by with on 1st 1st don 2nd contact telephone, Outcome of Date) attempt? contact!, attempt contact telephone, Outcome of Date) it is yes Mmm- No Mmm- |

Clinical Study Protocol: AMIC-003-CMD Time is 24 Hour clock

<sup>2</sup>Refers to either contact or attempt date and time Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Listing Status: DRAFT; SAS Program: Listing 16.11.sas


Listing 16.12.1 Listing of Adverse Events Post Procedure All Subjects Enrolled (N=xx)

| Outcome<br>End date | Recovere d/<br>Mmm-dd-<br>yyyy | Cont | Recovere d/<br>Mmm-dd-<br>yyyy | Cont |
|---|---|---|---|---|
| Serio<br>us/<br>Reaso<br>n | Š. | Yes/<br>Hospit<br>alizati<br>on | No | Yes/<br>Hospit<br>alizati |
| Relati<br>on-<br>ship<br>to<br>Devic | Not<br>Relate<br>d | Possi<br>bly<br>Relate<br>d | Unlik<br>ely<br>Relate<br>d | Relate<br>d |
| Relati<br>on-<br>ship to<br>Proce<br>dure | Possibl<br>y<br>Relate | Not<br>Relate<br>d | Relate | Unlike<br>ly<br>Relate<br>d |
| Action<br>Taken<br>(Subject | No | Yes | No | Yes |
| Action<br>Taken<br>(Procedure) | No Change | Interrupted | Change in<br>Parameters/<br>specify | Interrupted |
| Episode<br>Pattern | Single | Cont | Single | Con |
| Severity | Mild | Severe | Mild | Severe |
| Start<br>Date | Mmm-<br>dd-<br>yyyy | Mmm-<br>dd-<br>yyyy | Mmm-<br>dd-<br>yyyy | Mmm-<br>dd-<br>yyyy |
| Descriptio<br>n of<br>Event | Nausea | Chills | Other:<br>specify | Chills |
| AE<br>Number | | | | |
| Any<br>AEs? | Yes | Yes | Yes | Yes |
| Study<br>Site | BCW | BCW | BCW | KCI |
| Subje<br>ct ID | XXXXX | XXXXX | XXXXX | XXXXX |

Clinical Study Protocol: AMIC-003-CMD
Note: NA=Not Applicable; UNK=Unknown; ND=Not Done
AEs=adverse event
Listing Status: DRAFT; SAS Program: Listing 16.12.1.sas


Listing 16.12.2
Listing of MedDRA Coded Adverse Events Post-Procedure
All Subjects Enrolled (N=xx)

Clinical Study Protocol: AMIC-003-CMD
Note: NA=Not Applicable; UNK=Unknown; ND=Not Done
Listing Status: DRAFT; SAS Program: Listing 16.12.2.sas


Listing of Input Parameters - Pre-Procedure All Subjects Enrolled (N=xx)

| FCR (%) | End Hct<br>(%) | Depletion<br>Hct <sup>1</sup><br>(%) | Replacement<br>Volume<br>(mL) | Fluid<br>Balance<br>(mL) | AC<br>Ratio<br>(X:1) | Start Prime Hct (%) | End Prime Hct (%) |
|---|---|---|---|---|---|---|---|
| XX | XX | XX | XX | XX | XX | XX | XX |
| XX | XX | XX | XX | XX | XX | XX | XX |
| XX | XX | XX | XX | XX | XX | XX | XX |

<sup>1</sup>Applicable for Depletion/Exchange Procedures Note: NA=Not Applicable; UNK=Unknown; ND=Not Done FCR=fraction of cells remaining, AC=anticoagulant; Hct=hematocrit Listing Status: DRAFT; SAS Program: Listing 16.13.1.sas


Listing of Estimator Parameters Pre-Procedure All Subjects Enrolled (N=xx)

| Depletion Red Cell Volume <sup>1</sup> (mL) | XX | xx | XX |
|---------------------------------------------|-------|-------|-------|
| Other<br>Replacement<br>Fluid<br>(mL) | XX | XX | XX |
| AC<br>Used<br>(mL) | XX | XX | XX |
| AC to<br>Subject<br>(mL) | XX | XX | XX |
| Procedure<br>Time<br>(minutes) | XX | XX | XX |
| Whole Blood<br>Flow Rate<br>(mL/min) | XX | XX | XX |
| Subject<br>ID | XXXXX | XXXXX | XXXXX |

<sup>1</sup>Applicable for Depletion/Exchange Procedures Note: NA=Not Applicable; UNK=Unknown; ND=Not Done AC=anticoagulant; Hct=hematocrit Listing Status: DRAFT; SAS Program: Listing 16.13.1.sas


Listing 16.13.3 Listing of Input Procedure Parameters All Subjects Enrolled (N=xx)

| Subject Subjec Was Average Was Total ID t Hct Value Replacemen Value Blood (%) changed t Fluid Hct changed Volum during (%) during e procedure ? | WasAverageWasValueReplacemenValuechangedt Fluid Hctchangedduring(%)duringprocedure?retf V.?re | Was Value changed during procedu re | | Total<br>Blood<br>Volum<br>e<br>(mL) | | Was Value changed during procedure? | Max<br>Whole<br>Blood<br>Flow<br>Rate<br>(mL/mi | Was Value changed during procedure? | Citrate<br>Infusion<br>Rate<br>(mg/kg/<br>min) | Was Value changed during procedure? If Yes, |
|---|---|---|---|---|---|---|---|---|---|---|
| Final<br>Value | Final value | | | If Yes,<br>Final<br>Value | | Value | | Value | | Fillal Value |
| xx Yes, xx xx | | XX | | Yes, xx | XXX | Yes ,xx | XX | Yes, xx | XX | Yes, xx |
| xx Yes, xx Y | XX | | Y | Yes, xx | XXX | Yes, xx | XX | Yes ,xx | XX | Yes, xx |
| xx No xx | | XX | | No | XXX | No | XX | No | XX | No |
| ١, | | ١, | | | | | | | | |

Clinical Study Protocol: AMIC-003-CMD
Note: NA=Not Applicable; UNK=Unknown; ND=Not Done
Hct=hematocrit; Max=maximum; RBC=red blood cell; WB=whole Blood
Listing Status: DRAFT; SAS Program: Listing 16.13.2.sas


 $Listing \ 16.14 \\ Listing \ of End \ of Depletion \ Phase \ Parameters^1$ All Subjects (N=xx)

| Subject | | Depletion | WB | Replacement | Replacement | Custom | Plasma | Procedure | AC | AC to | Saline to |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Balance | Het | Processed | Fluid | Fluid Saline | | Returned | Time | <b>Used</b> | Subject | Subject |
| | (mL) | (%) | (mL) | Albumin | Returned | Fluid | (mL) | (minutes) | (mL) | (mL) | (mL) |
| | | | | Returned | (mL) | | 8 | ę. | | | 8 |
| | | | | (mL) | 5 | | | | | | |
| XXXXX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| XXXXX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| XXXXX | XX | xx | XX | XX | XX | XX | XX | XX | XX | XX | XX |

<sup>1</sup>Applicable for Depletion/Exchange Procedures
Note: NA=Not Applicable; UNK=Unknown; ND=Not Done
AC=anticoagulant; Hct=hematocrit; WB=whole blood
Listing Status: DRAFT; SAS Program: Listing 16.14.sas

Listing 16.15.1 Listing of Procedure Results All Subjects Enrolled (N=xx)

<sup>1</sup>For calculated parameters refer to algorithm document (AD) Note: NA=Not Applicable; UNK=Unknown; ND=Not Done AC=anticoagulant; Hct=hematocrit; WB=whole blood Listing Status: DRAFT; SAS Program: Listing 16.15.1.sas


Listing 16.15.2 Listing of Procedure Results All Subjects Enrolled (N=xx)

| Subject ID | Saline to Subject (mL) | Replacement Fluid<br>Albumin Returned<br>(mL) | Replacement<br>Fluid RBC<br>Returned<br>(mL) | Replacement<br>Fluid Saline<br>Returned<br>(mL) <sup>1</sup> | Custom Replacement Fluid Returned (mL) <sup>1</sup> |
|---|---|---|---|---|---|
| XXXX | XX | XX | XX | XX | XX |
| XXXX | XX | XX | XX | XX | XX |
| XXXX | XX | XX | XX | XX | XX |
| XXXX | XX | XX | XX | XX | XX |
| | 20 000 000 | | | | |

Clinical Study Protocol: AMIC-003-CMD

Applicable for Depletion/Exchange procedures

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done
RBC=red blood cell

Listing Status: DRAFT; SAS Program: Listing 16.15.2.sas

All Subjects Enrolled (N=xx) Listing 16.16 Listing of Primary Endpoint

| Pre-Procedure<br>Hemoglobin S<br>(%) | Post-Procedure<br>Hemoglobin S<br>(%) | FCR <sup>1</sup> (%) | Actual FCR <sup>2</sup> (%) | Calculated A:T<br>FCR<br>Ratio <sup>2</sup> |
|---|---|---|---|---|
| XX.XX | XX.XX | XX.XX | XX.XX | XX.X |
| XX.XX | XX.XX | XX.XX | XX.XX | X.XX |
| XX.XX | XX.XX | XX.XX | XX.XX | X.XX |

Clinical Study Protocol: AMIC-003-CMD

<sup>1</sup>Fraction of Cells Remaining reported by AMICUS at end of procedure.

<sup>2</sup>For calculated parameters refer to algorithm document (AD)

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done

FCR=fraction of cells remaining Listing Status: DRAFT; SAS Program: Listing 16.16.sas

Listing 16.17.1 Listing of Secondary Endpoints<sup>1</sup> All Subjects Enrolled (N=xx)

| Subject Plasma Hb Delta (mg/dL) | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
|---|---|---|---|---|---|
| Subject<br>Platelet<br>Percent<br>Loss<br>(%) | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Subject RBC Percent Loss (%) | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Subject WBC Percent Loss (%) | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Target End Hct Accuracy (%) | XX.X | X.XX | XXX.X | XX.X | XX.X |
| Subject Depletion Plasma Hb Delta <sup>2</sup> (mg/dL) | XX.X | XX.X | XXX.X | XXX.X | XX.X |
| Subject Depletion Platelet Percent Loss <sup>2</sup> (%) | XXX.X | XX.X | XX.X | XX.X | XX.X |
| Subject Depletion RBC Percent Loss <sup>2</sup> (%) | XX.X | XXX.X | XX.X | XX.X | XX.X |
| Subject Depletion WBC Percent Loss² (%) | XX.X | xx.x | XX.X | XX.X | XX.X |
| Depletion Het Accuracy <sup>2</sup> (%) | xx.x | XX.X | XX.X | XX.X | XX.X |
| Subject<br>ID | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |

<sup>1</sup>For calculated parameters refer to algorithm document (AD) <sup>2</sup>Applicable for Depletion/Exchange procedures Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Hct=hematocrit; RBC=red blood cell; WBC=white blood cell

Listing Status: DRAFT; SAS Program: Listing 16.17.1.sas


Listing of Waste Material for Secondary Endpoints<sup>1</sup> All Subjects Enrolled (N=xx)

| Subject Depletion Exchange Phase Pha | L | 0 | | | | | |
|---|---|---|---|---|---|---|---|
| XX.X XX.X XX.X XX.X XX.X XX.X | Depletion E Phase Waste WBC Count (x10 <sup>10</sup> ) | Exchange Phase Waste WBC Count (x10 <sup>10</sup> ) | Depletion Phase Waste Platelet Count (x10 <sup>11</sup> ) | Exchange Phase Waste Platelet Count (x10 <sup>11</sup> ) | Waste<br>Material<br>Volume<br>(mL) | Waste<br>WBC<br>Count<br>(x10 <sup>10</sup> ) | Waste<br>Platelet<br>Count<br>(x10 <sup>11</sup> ) |
| XX.X XX.X XX.X XX.X | XX.X | XX.X | XX.X | XXXX.X | XX.X | XX.X | XXXX.X |
| XX.X XX.X | XX.X | XX.X | XX.X | XXXX.X | XX.X | XX.X | XXXX.X |
| | XX.X | XX.X | XX.X | XXXX.X | XX.X | XX.X | XXXX.X |
| XXXXX XX.X XX.X | XX.X | XX.X | XX.X | XXXX.X | XX.X | XX.X | XXXX.X |
| CXX X.XX X.XX | XX.X | X.XX | X.XX | XXXX.X | XX.X | XX.X | XXX.X |

<sup>1</sup>For calculated parameters refer to algorithm document (AD) Note: NA=Not Applicable; UNK=Unknown; ND=Not Done WBC=white blood cell Listing Status: DRAFT; SAS Program: Listing 16.17.2.sas


Listing 16.17.3 Listing of End Hematocrit All Subjects Enrolled (N=xx)

| Hct <sup>1</sup> De | Subject Fost- | | Target | Procedure | Subject Post- | Della |
|---|---|---|---|---|---|---|
| | Depletion Phase | End of Depletion | Exchange End | | Procedure | End of Exchange |
| (%) | Hct <sup>2</sup> | | Hct <sup>3</sup> | | Hct <sup>2</sup> | Het. |
| | (%) | (%) | (%) | (%) | (%) | (0/) |
| XX | XX | XX | XX | XX | XX | XX |
| XX | XX | XX | XX | XX | XX | XX |
| XX | XX | XX | XX | XX | XX | XX |
| XX | XX | XX | XX | XX | XX | XX |

<sup>1</sup>End Hct (%) results reported Post-Depletion Phase.

<sup>2</sup>Subject laboratory measured values

<sup>3</sup>Target Hct entered Pre-Procedure

<sup>4</sup>End Hct (%) results reported Post-Procedure

<sup>5</sup>For calculated parameters refer to the algorithm document (AD) Note: NA=Not Applicable; UNK=Unknown; ND=Not Done; Hct=hematocrit; Listing Status: DRAFT; SAS Program: Listing 16.17.3.sas

Listing 16.18
Listing of Replacement RBC Unit Parameters
All Subjects Enrolled (N=xx)

| Subject<br>ID | Subject Type of ID RBC Unit | Unit ID<br>Number | Date<br>Sample<br>Drawn | Time<br>Sample<br>Drawn | Hct (%) | Volume (mL) | Total<br>Volume<br>(mL) | ABO<br>Type/<br>Rh<br>Factor | Expiration<br>Date | Plasma<br>Hb<br>(mg/dL) | Confirma<br>tion of<br>Sickle<br>Trait<br>Negative | Confirma<br>tion of<br>Leukored<br>uction | Confirma tion of RH (D) Compatib |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | CPD | XX | Mmm-dd-<br>yyyy | hh:mm | XX | XX | XX | × | Mmm-dd-<br>yyyy | XX | Yes | Yes | Yes |
| XXXXX | Other | XX | Mmm-dd- | hh:mm | XX | XX | XX | XX | Mmm-dd-<br>yyyy | XX | No | No | Yes |
| XXXXX | Washed<br>RBCs | XX | Mmm-dd-<br>yyyy | hh:mm | XX | XX | XX | XX | Mmm-dd-<br>yyyy | XX | No | Yes | No |
| Clinical S | hidy Protoce | Clinical Study Protocol. AMIC-003-CMD | 3-CMD | | | | | | | | | | |

Clinical Study Protocol: AMIC-003-CMD
Note: NA=Not Applicable; UNK=Unknown; ND=Not Done

Hb=hemoglobin; Hct=hematocrit; RBC=red blood cell Listing Status: DRAFT; SAS Program: Listing 16.18.sas


Listing 16.19
Listing of Device Alarms
All Subjects Enrolled (N=xx)

| Subject ID | Did alarm(s) occur during the procedure? | If yes, record all alarms that occurred | Frequency (Occurrence per procedure) |
|---|---|---|---|
| | | | X |
| XXXXX | Yes | ACD Flow Problem | 4 |
| XXXXX | No | | |
| XXXXX | Yes | Blood Warmer Prime Flow | 2 |
| XXXXX | Yes | Empty Saline | 3 |

Clinical Study Protocol: AMIC-003-CMD
Note: NA=Not Applicable; UNK=Unknown; ND=Not Done
Listing Status: DRAFT; SAS Program: Listing 16.19.sas


 $\label{eq:listing_problem} Listing~16.20$   $\label{eq:listing_problem} Listing~of~Waste~Material - RBC~Depletion/Exchange~Procedures \\ All~Subjects~Enrolled~(N=xx)$ 

| | Hct<br>(%) | XX | XX | XX | XX | |
|---|---|---|---|---|---|---|
| | Total Platelet Count (x10 <sup>11</sup> ) <sup>1</sup> | XX.X | XX.X | XX.X | XX.X | |
| | Platele<br>t<br>Count<br>(x10 <sup>3</sup> /μ<br>L) | XX | XX | XX | XX | |
| ge Phase | Total WBC Count (x10 <sup>10</sup> ) <sup>1</sup> | XX.X | XX.X | XX.X | XX.X | |
| RBC Exchange Phase | WBC<br>Count<br>(x10 <sup>3</sup> /µL) | XX.X | XX.X | XX.X | XX.X | |
| | Volume(<br>mL) <sup>1</sup> | XX | XX | XX | XX | |
| | Tare<br>Weight<br>(g) | XXX | XXX | XXX | XXX | |
| | Gross<br>Weight<br>(g) | XXX | XXX | XXX | XXX | |
| | Hct<br>(%) | XX | XX | XX | XX | |
| | Total Platelet Count (x10 <sup>11</sup> ) <sup>1</sup> | XX.X | XX.X | XX.X | XX.X | |
| 0 | Platelet<br>Count<br>(x10 <sup>3</sup> /µL) | XX | XX | XX | XX | |
| RBC Depletion Phase | Total WBC Count (x10 <sup>10</sup> ) <sup>1</sup> | XX.X | XX.X | XX.X | XXX.X | |
| RBC Deple | WBC<br>Count<br>(x10³/μ<br>L) | XXX.X | XX.X | XX.X | X.X.X | |
| | Volume(<br>mL) <sup>1</sup> | XX | XX | XX | XX | 'MD |
| | Tare<br>Weigh<br>t<br>(g) | XX | XX | XX | XX | VIC-003-C |
| | Gross<br>Weight<br>(g) | XXX | XXX | XXX | xxx | Clinical Study Protocol: AMIC-003-CMF |
| | Subject<br>ID | XXXXX | XXXXX | XXXXX | XXXXX | Clinical Study |

Clinical Study Protocol: AMIC-003-CMD

1-For calculated parameters refer to algorithm document (AD)

Note: NA=Not Applicable; UNK=Unknown; ND=Not Done
Hct=hematocrit; RBC=red blood cell; WBC=white blood cell

Listing Status: DRAFT; SAS Program: Listing 16.20.sas


Listing of Waste Material - RBC Exchange All Subjects Enrolled (N=xx)

| Subject ID | Gross<br>Weight<br>(g) | Tare Weight (g) | Volume (mL) <sup>1</sup> | WBC<br>Count<br>(x10 <sup>3</sup> /µL) | Total WBC Count | Platelet<br>Count<br>(x10 <sup>3</sup> /μL) | Total Platelet Count | Hct<br>(%) |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XX | XXX.X | XX | XX | XX.X | XX | ( XX.X | XXX |
| XXXXX | XX | XX.X | XX | XX | XX.X | XX | XX.X | XXX |
| XXXXX | XX | XX.X | XX | XX | XX.X | XX | XX.X | XXX |
| XXXXX | XX | XX.X | XX | XX | XX.X | XX | X.XX | XXX |
| CAND COO DIAM 1 4 4 1 10 1 110 | A A A A A A A A A A A A A A A A A A A | CIVED COO D | | | | | | |

<sup>1</sup>For calculated parameters refer to algorithm document (AD) Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Hct=hematocrit; WBC=white blood cell Listing Status: DRAFT; SAS Program: Listing 16.21.sas


Listing 16.22 Listing of Protocol Deviation All Subjects Enrolled (N=xx)

| Yes No Yes Yes Yes Yes | | | |
|---|---|---|---|
| No<br>Yes<br>Yes | Mimm-dd-yyyy | Inclusion Criteria | Subject ≥ 6 years old |
| Yes No Yes Yes | Mmm-dd-yyyy | Exclusion Criteria | Subjects who are pregnant |
| No<br>Yes<br>Yes | Mmm-dd-yyyy | Sampling/<br>Testing<br>Issues | Sample<br>Lost/Broken/Mislabel<br>ed |
| Yes | Mmm-dd-yyyy | Procedure Related Issues | Incorrect Use |
| Yes | Mmm-dd-yyyy | Subject receives the wrong treatment or incorrect dose | Randomization |
| | Mmm-dd-yyyy | Informed consent issues (specify) | |
| WIMM- | Mmm-dd-yyyy | Follow-Up not performed | |
| xxxxx Yes Mmm- | Mmm-dd-yyyy | Follow-Up outside of window | |
| XXXXX No Mmm- | Mmm-dd-yyyy | Other | |

Clinical Study Protocol: AMIC-003-CMD Note: NA=Not Applicable; UNK=Unknown; ND=Not Done Listing Status: DRAFT; SAS Program: Listing 16.22.sas

